CLINICAL TRIAL: NCT00586339
Title: Evaluation of the Safety and Immunogenicity of GlaxoSmithKline Biologicals' HPV Vaccine 580299 (Cervarix) in Adult Human Immunodeficiency Virus (HIV) Infected Female Subjects
Brief Title: Safety and Immunogenicity of GlaxoSmithKline Biologicals' HPV Vaccine 580299 (Cervarix) in HIV Infected Females
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 107863
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Infections, Papillomavirus
Keywords: HPV; Human papillomavirus (HPV) vaccine; Human Immunodeficiency Virus (HIV); Cervical cancer; Papillomavirus
MeSH Terms: conditions — Papillomavirus Infections; Acquired Immunodeficiency Syndrome; Uterine Cervical Neoplasms | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- HIV+/Cervarix Group (Experimental): Human immunodeficiency virus positive (HIV+) female subjects who received 3 doses of Cervarix vaccine administrated by intramuscular injection into the deltoid region of the non-dominant arm, according to a 0, 1, 6-month schedule.
  Interventions: Biological: Cervarix
- HIV+/Aluminium Hydroxide Group (Active Comparator): Human immunodeficiency virus positive (HIV+) female subjects who received 3 doses of control Aluminium Hydroxide [Al(OH)3], administrated by intramuscular injection into the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: Placebo Control
- HIV-/Cervarix Group (Experimental): Human immunodeficiency virus negative (HIV-) subjects who received 3 doses of Cervarix vaccine administrated by intramuscular injection into the deltoid region of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: Cervarix

INTERVENTIONS:
Biological: Cervarix — Intramuscular injection, 3 doses
  Arms: HIV+/Cervarix Group; HIV-/Cervarix Group
Biological: Placebo Control — Intramuscular injection, 3 doses
  Arms: HIV+/Aluminium Hydroxide Group

SUMMARY:
Infection with human papillomavirus (HPV) has been clearly established as the central cause of cervical cancer. The current study is designed to evaluate the safety and immunogenicity of GlaxoSmithKline Biologicals' HPV vaccine 580299 in HIV infected adult females living in the Republic of South Africa. The study is double blinded, randomized for HIV positive subjects and open for HIV negative subjects. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol
* A female between, and including, 18 and 25 years of age at the time of the first vaccination.
* Written, signed or thumb-printed informed consent obtained from the subject prior to enrolment.
* Subjects willing to undergo HIV Voluntary Counseling and Testing (VCT) and willing to be informed of their HIV status.
* Subjects willing to provide place of residence and be visited at home.
* HIV seropositive subjects:

  1. Subjects must be HIV seropositive according to WHO case definition
  2. Subjects with WHO Clinical Stage 1 HIV-associated disease
  3. Subjects currently on antiretroviral therapy (ART) must be compliant to ART and have undetectable viral load
* HIV seronegative subjects: Subjects confirmed as HIV seronegative at the screening visit are eligible to participate in the HIV-/HPV group of the study.
* Non-virgin subjects must have a normal colposcopy at the screening visit.
* Non-virgin subjects must have a normal cervical cytology (Pap smear) or no greater than atypical squamous cells of undetermined significance (ASC-US) at the screening visit.
* All subjects must have a negative urine pregnancy test at the screening visit and at visit 1 (Day 0).
* Subjects must be of non-childbearing potential or, if of childbearing potential, must be abstinent or have used adequate contraceptive precautions for 30 days prior to vaccination, have a negative pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series.
* Subjects must have had no more than 6 life-time sexual partners prior to enrolment.
* Subjects must have one single intact cervix

Exclusion Criteria:

* Active tuberculosis (TB)
* Current TB prophylaxis or therapy.
* Anemia at the screening visit.
* increased creatinine at the screening visit.
* Increased hepatic enzym (ALT) at the screening visit
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine within 30 days preceding the first dose of study vaccine/control, or planned use during the entire study period (up to Month 12).
* Chronic administration of immunosuppressants or other immune-modifying drugs within 6 months prior to the first vaccine dose.
* Administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of study vaccine/control. Enrolment will be postponed until the subject is outside the specified window.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days before or 30 days after (i.e., Days 0-29) any dose of study vaccine.
* Previous vaccination against HPV, or planned administration of any HPV vaccine other than that foreseen by the study protocol during the study period (Month 0 to Month 12).
* previous administration of components of the investigational vaccine
* Cancer or autoimmune disease under treatment.
* Hypersensitivity to latex.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine/control.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory testing performed at the screening visit.
* History of any neurological disorders or seizures.
* Pregnant or breastfeeding female.
* A subject planning to become pregnant, likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the study period, up to two months after the last vaccine dose.
* Concurrently participating in another clinical study, at any time during the study period (up to Month 12), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Any medically diagnosed or suspected immunodeficient condition (other than HIV for HIV seropositive subjects), based on medical history, physical examination and/or laboratory tests results.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine/control or planned administration during the study period. Enrolment will be postponed until the subject is outside the specified window.
* Administration of trimethoprim/sulphamethoxazole within 7 days before the first dose of study vaccine/control, or planned administration of trimethoprim/sulphamethoxazole within 7 days after the first dose of study vaccine/control.
* Current drugs or alcohol abuse.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-01-17 (Actual); Primary Completion 2011-07-18 (Actual); Study Completion 2011-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Khayelitsha, South Africa

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=2198

REFERENCES:
- [Background] Denny L, Hendricks B, Gordon C, Thomas F, Hezareh M, Dobbelaere K, Durand C, Herve C, Descamps D. Safety and immunogenicity of the HPV-16/18 AS04-adjuvanted vaccine in HIV-positive women in South Africa: a partially-blind randomised placebo-controlled study. Vaccine. 2013 Nov 19;31(48):5745-53. doi: 10.1016/j.vaccine.2013.09.032. Epub 2013 Oct 1. PMID 24091311
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 107863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 107863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV+ subjects were randomised to receive either Cervarix or Aluminium Hydroxide vaccines; HIV- subjects were not randomised and all received Cervarix vaccine.
Pre-assignment Details: Enrollment was staggered as follows: 1) Enrollment of Human immunodeficiency virus positive (HIV+) subjects with cluster of differentiation 4 (CD4+) cell count >200 cells per cubic millimeter (cells/mm^3) and HIV negative (HIV-) subjects (up to 30 subjects) for blinded safety evaluation; 2) Enrollment of remaining HIV+/HIV- subjects.
Period: Overall Study
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Started | 61 | 59 | 30
Completed | 54 | 52 | 24
Not Completed | 7 | 7 | 6
Not completed — Withdrawal by Subject | 1 | 3 | 1
Not completed — Migrated/moved from study area | 3 | 2 | 4
Not completed — Lost to Follow-up | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group | Total
Number analyzed (Participants) | 61 | 59 | 30 | 150
Age, Continuous [Mean (Standard Deviation); unit: Years] | 21.6 (2.21) | 22.7 (1.70) | 21.3 (1.65) | 21.9 (1.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 59 | 30 | 150
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 61 | 59 | 30 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain and swelling. Any = occurrence of any solicited local regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 swelling = swelling spreading beyond 50 millimeters (mm) of injection site. Solicited local symptoms were assessed as related to the study vaccination.
Time Frame: Within 7 days after each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who had their symptom sheet filled in and for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 61 | 59 | 30
Participants
  Any Pain, Dose 1 | 46 | 18 | 19
  Grade 3 Pain, Dose 1 | 2 | 0 | 0
  Any Swelling, Dose 1 | 6 | 0 | 4
  Grade 3 Swelling, Dose 1 | 1 | 0 | 2
  Any Pain, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Pain, Dose 2 | 29 | 12 | 21
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Pain, Dose 2 | 0 | 0 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Swelling, Dose 2 | 5 | 0 | 8
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Swelling, Dose 2 | 0 | 0 | 2
  Any Pain, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Pain, Dose 3 | 27 | 6 | 19
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Pain, Dose 3 | 1 | 0 | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Swelling, Dose 3 | 12 | 2 | 3
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Swelling, Dose 3 | 0 | 0 | 1
  Any Pain, Across doses | 52 | 27 | 28
  Grade 3 Pain, Across doses | 3 | 0 | 1
  Any Swelling, Across doses | 19 | 2 | 12
  Grade 3 Swelling, Across doses | 1 | 0 | 4

2. Primary Outcome: Number of Subjects Reporting Any, Severe (Grade 3) and Related Solicited General Symptoms
Description: Solicited general symptoms assessed were arthralgia, fatigue, fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)], gastrointestinal, headache, myalgia, rash and urticaria. Any = occurrence of any solicited general symptom regardless of their intensity grade or relationship. Grade 3 Symptom = symptom that prevented normal activity. Grade 3 Urticaria = Urticaria distributed on at least 4 body areas. Related = symptom assessed by the investigator as causally related to the vaccination.
Time Frame: Within 7 days after each dose and across doses
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 61 | 59 | 30
Participants
  Any Arthralgia, Dose 1 | 3 | 4 | 2
  Grade 3 Arthralgia, Dose 1 | 0 | 0 | 0
  Related Arthralgia, Dose 1 | 1 | 1 | 2
  Any Fatigue, Dose 1 | 12 | 13 | 7
  Grade 3 Fatigue, Dose 1 | 0 | 1 | 0
  Related Fatigue, Dose 1 | 9 | 9 | 5
  Any Fever, Dose 1 | 1 | 2 | 0
  Grade 3 Fever, Dose 1 | 0 | 1 | 0
  Related Fever, Dose 1 | 0 | 0 | 0
  Any Gastrointestinal, Dose 1 | 5 | 7 | 9
  Grade 3 Gastrointestinal, Dose 1 | 0 | 0 | 0
  Related Gastrointestinal, Dose 1 | 2 | 2 | 2
  Any Headache, Dose 1 | 13 | 16 | 11
  Grade 3 Headache, Dose 1 | 0 | 0 | 0
  Related Headache, Dose 1 | 5 | 4 | 1
  Any Myalgia, Dose 1 | 2 | 1 | 4
  Grade 3 Myalgia, Dose 1 | 0 | 0 | 0
  Related Myalgia, Dose 1 | 1 | 1 | 3
  Any Rash, Dose 1 | 0 | 2 | 0
  Grade 3 Rash, Dose 1 | 0 | 0 | 0
  Related Rash, Dose 1 | 0 | 1 | 0
  Any Urticaria, Dose 1 | 0 | 0 | 0
  Grade 3 Urticaria, Dose 1 | 0 | 0 | 0
  Related Urticaria, Dose 1 | 0 | 0 | 0
  Any Arthralgia, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Arthralgia, Dose 2 | 0 | 0 | 0
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Arthralgia, Dose 2 | 0 | 0 | 0
  Related Arthralgia, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Related Arthralgia, Dose 2 | 0 | 0 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Fatigue, Dose 2 | 4 | 6 | 4
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Fatigue, Dose 2 | 0 | 0 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Related Fatigue, Dose 2 | 4 | 4 | 4
  Any Fever, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Fever, Dose 2 | 0 | 0 | 0
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Fever, Dose 2 | 0 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Related Fever, Dose 2 | 0 | 0 | 0
  Any Gastrointestinal, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Gastrointestinal, Dose 2 | 10 | 2 | 4
  Grade 3 Gastrointestinal, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Gastrointestinal, Dose 2 | 1 | 0 | 0
  Related Gastrointestinal, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Related Gastrointestinal, Dose 2 | 3 | 1 | 0
  Any Headache, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Headache, Dose 2 | 11 | 9 | 4
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Headache, Dose 2 | 0 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Related Headache, Dose 2 | 5 | 2 | 1
  Any Myalgia, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Myalgia, Dose 2 | 0 | 1 | 3
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Myalgia, Dose 2 | 0 | 0 | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Related Myalgia, Dose 2 | 0 | 1 | 3
  Any Rash, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Rash, Dose 2 | 0 | 0 | 1
  Grade 3 Rash, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Rash, Dose 2 | 0 | 0 | 0
  Related Rash, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Related Rash, Dose 2 | 0 | 0 | 0
  Any Urticaria, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Any Urticaria, Dose 2 | 0 | 0 | 0
  Grade 3 Urticaria, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Grade 3 Urticaria, Dose 2 | 0 | 0 | 0
  Related Urticaria, Dose 2: number analyzed (Participants) | 53 | 51 | 29
  Related Urticaria, Dose 2 | 0 | 0 | 0
  Any Arthralgia, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Arthralgia, Dose 3 | 1 | 0 | 0
  Grade 3 Arthralgia, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Arthralgia, Dose 3 | 0 | 0 | 0
  Related Arthralgia, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Related Arthralgia, Dose 3 | 1 | 0 | 0
  Any Fatigue, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Fatigue, Dose 3 | 4 | 1 | 4
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Fatigue, Dose 3 | 0 | 0 | 0
  Related Fatigue, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Related Fatigue, Dose 3 | 4 | 1 | 4
  Any Fever, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Fever, Dose 3 | 1 | 1 | 2
  Grade 3 Fever, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Fever, Dose 3 | 0 | 0 | 0
  Related Fever, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Related Fever, Dose 3 | 1 | 0 | 0
  Any Gastrointestinal, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Gastrointestinal, Dose 3 | 3 | 2 | 6
  Grade 3 Gastrointestinal, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Gastrointestinal, Dose 3 | 0 | 0 | 0
  Related Gastrointestinal, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Related Gastrointestinal, Dose 3 | 1 | 0 | 3
  Any Headache, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Headache, Dose 3 | 2 | 7 | 6
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Headache, Dose 3 | 0 | 0 | 0
  Related Headache, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Related Headache, Dose 3 | 1 | 3 | 2
  Any Myalgia, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Myalgia, Dose 3 | 1 | 1 | 1
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Myalgia, Dose 3 | 0 | 0 | 0
  Related Myalgia, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Related Myalgia, Dose 3 | 1 | 1 | 1
  Any Rash, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Rash, Dose 3 | 1 | 0 | 0
  Grade 3 Rash, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Rash, Dose 3 | 0 | 0 | 0
  Related Rash, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Related Rash, Dose 3 | 0 | 0 | 0
  Any Urticaria, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Any Urticaria, Dose 3 | 0 | 0 | 0
  Grade 3 Urticaria, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Grade 3 Urticaria, Dose 3 | 0 | 0 | 0
  Related Urticaria, Dose 3: number analyzed (Participants) | 48 | 44 | 26
  Related Urticaria, Dose 3 | 0 | 0 | 0
  Any Arthralgia, Across doses | 4 | 4 | 2
  Grade 3 Arthralgia, Across doses | 0 | 0 | 0
  Related Arthralgia, Across doses | 2 | 1 | 2
  Any Fatigue, Across doses | 18 | 16 | 8
  Grade 3 Fatigue, Across doses | 0 | 1 | 0
  Related Fatigue, Across doses | 15 | 12 | 7
  Any Fever, Across doses | 2 | 3 | 2
  Grade 3 Fever, Across doses | 0 | 1 | 0
  Related Fever, Across doses | 1 | 0 | 0
  Any Gastrointestinal, Across doses | 15 | 11 | 13
  Grade 3 Gastrointestinal, Across doses | 1 | 0 | 0
  Related Gastrointestinal, Across doses | 5 | 3 | 4
  Any Headache, Across doses | 23 | 26 | 16
  Grade 3 Headache, Across doses | 0 | 0 | 0
  Related Headache, Across doses | 10 | 9 | 3
  Any Myalgia, Across doses | 3 | 3 | 7
  Grade 3 Myalgia, Across doses | 0 | 0 | 0
  Related Myalgia, Across doses | 2 | 3 | 7
  Any Rash, Across doses | 1 | 2 | 1
  Grade 3 Rash, Across doses | 0 | 0 | 0
  Related Rash, Across doses | 0 | 1 | 0
  Any Urticaria, Across doses | 0 | 0 | 0
  Grade 3 Urticaria, Across doses | 0 | 0 | 0
  Related Urticaria, Across doses | 0 | 0 | 0

3. Primary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Symptoms
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within 30 days after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 61 | 59 | 30
Participants
  Any unsolicited AE(s) | 53 | 46 | 26
  Grade 3 unsolicited AE(s) | 1 | 1 | 0
  Related unsolicited AE(s) | 16 | 3 | 7

4. Primary Outcome: Number of Subjects With Medically Significant Conditions (MSCs) From Day 0 up to Month 7
Description: Medically significant conditions (MSCs) were collected regardless of causal relationship to vaccination and intensity. Medically significant conditions were defined as adverse events (AEs) prompting emergency room or physician visits that were not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or serious adverse events (SAEs) that were not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From Day 0 up to Month 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 61 | 59 | 30
Participants | 18 | 21 | 5

5. Primary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs) From Day 0 up to Month 7
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 up to Month 7
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 61 | 59 | 30
Participants | 3 | 2 | 1

6. Primary Outcome: Number of Subjects With Pregnancies and Outcomes of Reported Pregnancies From Day 0 up to Month 7
Description: The subjects with confirmed pregnancies were followed up to determine the outcomes of the reported pregnancies. The outcome of the reported pregnancy was a live infant with no apparent congenital anomaly.
Time Frame: From Day 0 up to Month 7
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who reported pregnancies and outcomes of reported pregnancies.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 0 | 1 | 0
Participants |  | 1 |

7. Primary Outcome: Number of Subjects Reporting SAEs From Day 0 up to Month 12
Description: as for outcome 5
Time Frame: From Day 0 up to Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 61 | 59 | 30
Participants | 3 | 2 | 1

8. Primary Outcome: Number of Subjects With MSCs From Day 0 up to Month 12
Description: MSCs were collected regardless of causal relationship to vaccination and intensity. Medically significant conditions were defined as adverse events (AEs) prompting emergency room or physician visits that were not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or serious adverse events (SAEs) that were not related to common diseases. Common diseases include upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervico-vaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From Day 0 up to Month 12
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 61 | 59 | 30
Participants | 19 | 21 | 5

9. Primary Outcome: Number of Subjects With Pregnancies and Outcomes of Reported Pregnancies From Day 0 up to Month 12
Description: as for outcome 6
Time Frame: From Day 0 up to Month 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 0 | 1 | 0
Participants |  | 1 |

10. Primary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Red Blood Cells and Platelets Parameters at Day 7 and at Months 1, 2, 4, 6 and 7
Description: Haematological laboratory parameters assessed were red blood cells (RBC) and platelets (PLA). For each parameter and by pre-vaccination status, it was assessed whether the post-vaccination values of the parameter were above, below or in the normal range (missing values are also indicated).
Time Frame: At Day 7 and at Months 1, 2, 4, 6 and 7
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom assay results were available at the considered time points.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 56 | 55 | 29
Participants
  RBC [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 15 | 14 | 15
  RBC [pre-vacc Normal; post-vacc Normal] Day 7 | 14 | 12 | 15
  RBC [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 15 | 14 | 15
  RBC [pre-vacc Normal; post-vacc Below] Day 7 | 1 | 2 | 0
  RBC [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 15 | 14 | 15
  RBC [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 15 | 14 | 15
  RBC [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Normal] Month 1: number analyzed (Participants) | 51 | 48 | 29
  RBC [pre-vacc Normal; post-vacc Normal] Month 1 | 46 | 44 | 25
  RBC [pre-vacc Normal; post-vacc Below] Month 1: number analyzed (Participants) | 51 | 48 | 29
  RBC [pre-vacc Normal; post-vacc Below] Month 1 | 5 | 4 | 4
  RBC [pre-vacc Normal; post-vacc Above] Month 1: number analyzed (Participants) | 51 | 48 | 29
  RBC [pre-vacc Normal; post-vacc Above] Month 1 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Missing] Month 1: number analyzed (Participants) | 51 | 48 | 29
  RBC [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 49 | 48 | 28
  RBC [pre-vacc Normal; post-vacc Normal] Month 2 | 44 | 45 | 28
  RBC [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 49 | 48 | 28
  RBC [pre-vacc Normal; post-vacc Below] Month 2 | 5 | 3 | 0
  RBC [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 49 | 48 | 28
  RBC [pre-vacc Normal; post-vacc Above] Month 2 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 49 | 48 | 28
  RBC [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 49 | 46 | 26
  RBC [pre-vacc Normal; post-vacc Normal] Month 4 | 43 | 40 | 25
  RBC [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 49 | 46 | 26
  RBC [pre-vacc Normal; post-vacc Below] Month 4 | 6 | 6 | 1
  RBC [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 49 | 46 | 26
  RBC [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 49 | 46 | 26
  RBC [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 49 | 45 | 26
  RBC [pre-vacc Normal; post-vacc Normal] Month 6 | 40 | 40 | 25
  RBC [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 49 | 45 | 26
  RBC [pre-vacc Normal; post-vacc Below] Month 6 | 9 | 5 | 1
  RBC [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 49 | 45 | 26
  RBC [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 49 | 45 | 26
  RBC [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 48 | 45 | 25
  RBC [pre-vacc Normal; post-vacc Normal] Month 7 | 43 | 37 | 24
  RBC [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 48 | 45 | 25
  RBC [pre-vacc Normal; post-vacc Below] Month 7 | 5 | 8 | 1
  RBC [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 48 | 45 | 25
  RBC [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 48 | 45 | 25
  RBC [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Normal] Day 7: number analyzed (Participants) | 0 | 1 | 0
  RBC [pre-vacc Low; post-vacc Normal] Day 7 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Below] Day 7: number analyzed (Participants) | 0 | 1 | 0
  RBC [pre-vacc Low; post-vacc Below] Day 7 | 0 | 1 | 0
  RBC [pre-vacc Low; post-vacc Above] Day 7: number analyzed (Participants) | 0 | 1 | 0
  RBC [pre-vacc Low; post-vacc Above] Day 7 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Missing] Day 7: number analyzed (Participants) | 0 | 1 | 0
  RBC [pre-vacc Low; post-vacc Missing] Day 7 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 9 | 9 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 1 | 4 | 4 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 9 | 9 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 1 | 5 | 5 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 9 | 9 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 9 | 9 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 9 | 9 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 2 | 3 | 1 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 9 | 9 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 2 | 6 | 8 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 9 | 9 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 9 | 9 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 8 | 8 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 4 | 4 | 4 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 8 | 8 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 4 | 4 | 4 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 8 | 8 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 8 | 8 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 8 | 9 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 6 | 3 | 4 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 8 | 9 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 6 | 5 | 5 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 8 | 9 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 8 | 9 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 8 | 8 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 7 | 2 | 4 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 8 | 8 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 7 | 6 | 4 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 8 | 8 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 8 | 8 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 13 | 14 | 15
  PLA [pre-vacc Normal; post-vacc Normal] Day 7 | 13 | 14 | 15
  PLA [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 13 | 14 | 15
  PLA [pre-vacc Normal; post-vacc Below] Day 7 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 13 | 14 | 15
  PLA [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 13 | 14 | 15
  PLA [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Normal] Month 1 | 56 | 54 | 29
  PLA [pre-vacc Normal; post-vacc Below] Month 1 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Above] Month 1 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 1 | 0
  PLA [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 54 | 55 | 28
  PLA [pre-vacc Normal; post-vacc Normal] Month 2 | 51 | 54 | 28
  PLA [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 54 | 55 | 28
  PLA [pre-vacc Normal; post-vacc Below] Month 2 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 54 | 55 | 28
  PLA [pre-vacc Normal; post-vacc Above] Month 2 | 2 | 1 | 0
  PLA [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 54 | 55 | 28
  PLA [pre-vacc Normal; post-vacc Missing] Month 2 | 1 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 53 | 52 | 26
  PLA [pre-vacc Normal; post-vacc Normal] Month 4 | 52 | 51 | 26
  PLA [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 53 | 52 | 26
  PLA [pre-vacc Normal; post-vacc Below] Month 4 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 53 | 52 | 26
  PLA [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 1 | 0
  PLA [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 53 | 52 | 26
  PLA [pre-vacc Normal; post-vacc Missing] Month 4 | 1 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 53 | 52 | 26
  PLA [pre-vacc Normal; post-vacc Normal] Month 6 | 53 | 52 | 26
  PLA [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 53 | 52 | 26
  PLA [pre-vacc Normal; post-vacc Below] Month 6 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 53 | 52 | 26
  PLA [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 53 | 52 | 26
  PLA [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 52 | 51 | 25
  PLA [pre-vacc Normal; post-vacc Normal] Month 7 | 51 | 50 | 25
  PLA [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 52 | 51 | 25
  PLA [pre-vacc Normal; post-vacc Below] Month 7 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 52 | 51 | 25
  PLA [pre-vacc Normal; post-vacc Above] Month 7 | 1 | 1 | 0
  PLA [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 52 | 51 | 25
  PLA [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 1 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 1 | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 2 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 2 | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 4 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 4 | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 6 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 6 | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 7 | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 7 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Normal] Day 7: number analyzed (Participants) | 2 | 1 | 0
  PLA [pre-vacc High; post-vacc Normal] Day 7 | 0 | 1 | 0
  PLA [pre-vacc High; post-vacc Below] Day 7: number analyzed (Participants) | 2 | 1 | 0
  PLA [pre-vacc High; post-vacc Below] Day 7 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Above] Day 7: number analyzed (Participants) | 2 | 1 | 0
  PLA [pre-vacc High; post-vacc Above] Day 7 | 2 | 0 | 0
  PLA [pre-vacc High; post-vacc Missing] Day 7: number analyzed (Participants) | 2 | 1 | 0
  PLA [pre-vacc High; post-vacc Missing] Day 7 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 1: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 1 | 1 | 0 | 0
  PLA [pre-vacc High; post-vacc Below] Month 1: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 1 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Above] Month 1: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Above] Month 1 | 2 | 2 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 1: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 1 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 2: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 2 | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 2: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 2 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Above] Month 2: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Above] Month 2 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 2: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 2 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 4: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 4 | 2 | 1 | 0
  PLA [pre-vacc High; post-vacc Below] Month 4: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 4 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Above] Month 4: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Above] Month 4 | 1 | 1 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 4: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 4 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 6: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 6 | 3 | 1 | 0
  PLA [pre-vacc High; post-vacc Below] Month 6: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 6 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Above] Month 6: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Above] Month 6 | 0 | 1 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 6: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 6 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 7: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 7 | 2 | 1 | 0
  PLA [pre-vacc High; post-vacc Below] Month 7: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 7 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Above] Month 7: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Above] Month 7 | 1 | 1 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 7: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 7 | 0 | 0 | 0

11. Primary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in White Blood Cells and Neutrophils Parameters at Day 7 and Months 1, 2, 4, 6 and 7
Description: Haematological laboratory parameters assessed were white blood cells (WBC) and neutrophils (NEU). For each parameter and by pre-vaccination status, it was assessed whether the post-vaccination values of the parameter were above, below or in the normal range (missing values are also indicated).
Time Frame: At Day 7 and Months 1, 2, 4, 6 and 7
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 48 | 50 | 26
Participants
  WBC [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 13 | 14 | 13
  WBC [pre-vacc Normal; post-vacc Normal] Day 7 | 9 | 12 | 12
  WBC [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 13 | 14 | 13
  WBC [pre-vacc Normal; post-vacc Below] Day 7 | 4 | 2 | 1
  WBC [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 13 | 14 | 13
  WBC [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 13 | 14 | 13
  WBC [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Normal] Month 1: number analyzed (Participants) | 46 | 49 | 26
  WBC [pre-vacc Normal; post-vacc Normal] Month 1 | 39 | 43 | 23
  WBC [pre-vacc Normal; post-vacc Below] Month 1: number analyzed (Participants) | 46 | 49 | 26
  WBC [pre-vacc Normal; post-vacc Below] Month 1 | 7 | 6 | 3
  WBC [pre-vacc Normal; post-vacc Above] Month 1: number analyzed (Participants) | 46 | 49 | 26
  WBC [pre-vacc Normal; post-vacc Above] Month 1 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Missing] Month 1: number analyzed (Participants) | 46 | 49 | 26
  WBC [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 44 | 50 | 26
  WBC [pre-vacc Normal; post-vacc Normal] Month 2 | 38 | 41 | 24
  WBC [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 44 | 50 | 26
  WBC [pre-vacc Normal; post-vacc Below] Month 2 | 6 | 9 | 2
  WBC [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 44 | 50 | 26
  WBC [pre-vacc Normal; post-vacc Above] Month 2 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 44 | 50 | 26
  WBC [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 43 | 48 | 24
  WBC [pre-vacc Normal; post-vacc Normal] Month 4 | 37 | 41 | 22
  WBC [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 43 | 48 | 24
  WBC [pre-vacc Normal; post-vacc Below] Month 4 | 6 | 7 | 2
  WBC [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 43 | 48 | 24
  WBC [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 43 | 48 | 24
  WBC [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 43 | 46 | 24
  WBC [pre-vacc Normal; post-vacc Normal] Month 6 | 35 | 38 | 21
  WBC [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 43 | 46 | 24
  WBC [pre-vacc Normal; post-vacc Below] Month 6 | 8 | 8 | 2
  WBC [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 43 | 46 | 24
  WBC [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 1
  WBC [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 43 | 46 | 24
  WBC [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 42 | 46 | 23
  WBC [pre-vacc Normal; post-vacc Normal] Month 7 | 34 | 38 | 21
  WBC [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 42 | 46 | 23
  WBC [pre-vacc Normal; post-vacc Below] Month 7 | 8 | 8 | 2
  WBC [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 42 | 46 | 23
  WBC [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 42 | 46 | 23
  WBC [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Normal] Day 7: number analyzed (Participants) | 2 | 1 | 2
  WBC [pre-vacc Low; post-vacc Normal] Day 7 | 1 | 1 | 1
  WBC [pre-vacc Low; post-vacc Below] Day 7: number analyzed (Participants) | 2 | 1 | 2
  WBC [pre-vacc Low; post-vacc Below] Day 7 | 1 | 0 | 1
  WBC [pre-vacc Low; post-vacc Above] Day 7: number analyzed (Participants) | 2 | 1 | 2
  WBC [pre-vacc Low; post-vacc Above] Day 7 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Missing] Day 7: number analyzed (Participants) | 2 | 1 | 2
  WBC [pre-vacc Low; post-vacc Missing] Day 7 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 14 | 8 | 3
  WBC [pre-vacc Low; post-vacc Normal] Month 1 | 9 | 5 | 2
  WBC [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 14 | 8 | 3
  WBC [pre-vacc Low; post-vacc Below] Month 1 | 5 | 3 | 1
  WBC [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 14 | 8 | 3
  WBC [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 14 | 8 | 3
  WBC [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 14 | 7 | 2
  WBC [pre-vacc Low; post-vacc Normal] Month 2 | 10 | 5 | 0
  WBC [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 14 | 7 | 2
  WBC [pre-vacc Low; post-vacc Below] Month 2 | 4 | 2 | 2
  WBC [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 14 | 7 | 2
  WBC [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 14 | 7 | 2
  WBC [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 14 | 6 | 2
  WBC [pre-vacc Low; post-vacc Normal] Month 4 | 8 | 2 | 1
  WBC [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 14 | 6 | 2
  WBC [pre-vacc Low; post-vacc Below] Month 4 | 6 | 4 | 1
  WBC [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 14 | 6 | 2
  WBC [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 14 | 6 | 2
  WBC [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 14 | 8 | 2
  WBC [pre-vacc Low; post-vacc Normal] Month 6 | 6 | 5 | 0
  WBC [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 14 | 8 | 2
  WBC [pre-vacc Low; post-vacc Below] Month 6 | 8 | 3 | 2
  WBC [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 14 | 8 | 2
  WBC [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 14 | 8 | 2
  WBC [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 14 | 7 | 2
  WBC [pre-vacc Low; post-vacc Normal] Month 7 | 6 | 3 | 1
  WBC [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 14 | 7 | 2
  WBC [pre-vacc Low; post-vacc Below] Month 7 | 8 | 4 | 1
  WBC [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 14 | 7 | 2
  WBC [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 14 | 7 | 2
  WBC [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 13 | 14 | 13
  NEU [pre-vacc Normal; post-vacc Normal] Day 7 | 9 | 11 | 12
  NEU [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 13 | 14 | 13
  NEU [pre-vacc Normal; post-vacc Below] Day 7 | 4 | 3 | 1
  NEU [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 13 | 14 | 13
  NEU [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 13 | 14 | 13
  NEU [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Normal] Month 1: number analyzed (Participants) | 48 | 41 | 25
  NEU [pre-vacc Normal; post-vacc Normal] Month 1 | 36 | 36 | 21
  NEU [pre-vacc Normal; post-vacc Below] Month 1: number analyzed (Participants) | 48 | 41 | 25
  NEU [pre-vacc Normal; post-vacc Below] Month 1 | 11 | 5 | 4
  NEU [pre-vacc Normal; post-vacc Above] Month 1: number analyzed (Participants) | 48 | 41 | 25
  NEU [pre-vacc Normal; post-vacc Above] Month 1 | 1 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Missing] Month 1: number analyzed (Participants) | 48 | 41 | 25
  NEU [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 46 | 42 | 25
  NEU [pre-vacc Normal; post-vacc Normal] Month 2 | 38 | 35 | 22
  NEU [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 46 | 42 | 25
  NEU [pre-vacc Normal; post-vacc Below] Month 2 | 8 | 6 | 3
  NEU [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 46 | 42 | 25
  NEU [pre-vacc Normal; post-vacc Above] Month 2 | 0 | 1 | 0
  NEU [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 46 | 42 | 25
  NEU [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 45 | 40 | 23
  NEU [pre-vacc Normal; post-vacc Normal] Month 4 | 36 | 30 | 19
  NEU [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 45 | 40 | 23
  NEU [pre-vacc Normal; post-vacc Below] Month 4 | 9 | 10 | 4
  NEU [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 45 | 40 | 23
  NEU [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 45 | 40 | 23
  NEU [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 45 | 38 | 23
  NEU [pre-vacc Normal; post-vacc Normal] Month 6 | 33 | 33 | 19
  NEU [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 45 | 38 | 23
  NEU [pre-vacc Normal; post-vacc Below] Month 6 | 12 | 5 | 4
  NEU [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 45 | 38 | 23
  NEU [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 45 | 38 | 23
  NEU [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 44 | 38 | 22
  NEU [pre-vacc Normal; post-vacc Normal] Month 7 | 35 | 32 | 18
  NEU [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 44 | 38 | 22
  NEU [pre-vacc Normal; post-vacc Below] Month 7 | 9 | 6 | 4
  NEU [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 44 | 38 | 22
  NEU [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 44 | 38 | 22
  NEU [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Normal] Day 7: number analyzed (Participants) | 2 | 1 | 2
  NEU [pre-vacc Low; post-vacc Normal] Day 7 | 0 | 1 | 0
  NEU [pre-vacc Low; post-vacc Below] Day 7: number analyzed (Participants) | 2 | 1 | 2
  NEU [pre-vacc Low; post-vacc Below] Day 7 | 2 | 0 | 2
  NEU [pre-vacc Low; post-vacc Above] Day 7: number analyzed (Participants) | 2 | 1 | 2
  NEU [pre-vacc Low; post-vacc Above] Day 7 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Missing] Day 7: number analyzed (Participants) | 2 | 1 | 2
  NEU [pre-vacc Low; post-vacc Missing] Day 7 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 12 | 16 | 4
  NEU [pre-vacc Low; post-vacc Normal] Month 1 | 7 | 6 | 1
  NEU [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 12 | 16 | 4
  NEU [pre-vacc Low; post-vacc Below] Month 1 | 5 | 10 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 12 | 16 | 4
  NEU [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 12 | 16 | 4
  NEU [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 12 | 15 | 3
  NEU [pre-vacc Low; post-vacc Normal] Month 2 | 6 | 7 | 0
  NEU [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 12 | 15 | 3
  NEU [pre-vacc Low; post-vacc Below] Month 2 | 6 | 8 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 12 | 15 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 12 | 15 | 3
  NEU [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Normal] Month 4 | 6 | 7 | 1
  NEU [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Below] Month 4 | 6 | 7 | 2
  NEU [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 12 | 16 | 3
  NEU [pre-vacc Low; post-vacc Normal] Month 6 | 5 | 6 | 0
  NEU [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 12 | 16 | 3
  NEU [pre-vacc Low; post-vacc Below] Month 6 | 7 | 10 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 12 | 16 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 12 | 16 | 3
  NEU [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 12 | 15 | 3
  NEU [pre-vacc Low; post-vacc Normal] Month 7 | 5 | 6 | 0
  NEU [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 12 | 15 | 3
  NEU [pre-vacc Low; post-vacc Below] Month 7 | 7 | 9 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 12 | 15 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 12 | 15 | 3
  NEU [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0

12. Primary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Lymphocytes and Monocytes Parameters at Day 7 and Months 1, 2, 4, 6 and 7
Description: Haematological laboratory parameters assessed were lymphocytes (LYM) and monocytes (MON). For each parameter and by pre-vaccination status, it was assessed whether the post-vaccination values of the parameter were above, below or in the normal range (missing values are also indicated).
Time Frame: At Day 7 and at Months 1, 2, 4, 6 and 7
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 57 | 56 | 29
Participants
  LYM [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 12 | 14 | 14
  LYM [pre-vacc Normal; post-vacc Normal] Day 7 | 12 | 14 | 14
  LYM [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 12 | 14 | 14
  LYM [pre-vacc Normal; post-vacc Below] Day 7 | 0 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 12 | 14 | 14
  LYM [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 12 | 14 | 14
  LYM [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Normal] Month 1: number analyzed (Participants) | 54 | 56 | 27
  LYM [pre-vacc Normal; post-vacc Normal] Month 1 | 52 | 55 | 27
  LYM [pre-vacc Normal; post-vacc Below] Month 1: number analyzed (Participants) | 54 | 56 | 27
  LYM [pre-vacc Normal; post-vacc Below] Month 1 | 2 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Above] Month 1: number analyzed (Participants) | 54 | 56 | 27
  LYM [pre-vacc Normal; post-vacc Above] Month 1 | 0 | 1 | 0
  LYM [pre-vacc Normal; post-vacc Missing] Month 1: number analyzed (Participants) | 54 | 56 | 27
  LYM [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 52 | 56 | 26
  LYM [pre-vacc Normal; post-vacc Normal] Month 2 | 50 | 54 | 26
  LYM [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 52 | 56 | 26
  LYM [pre-vacc Normal; post-vacc Below] Month 2 | 1 | 2 | 0
  LYM [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 52 | 56 | 26
  LYM [pre-vacc Normal; post-vacc Above] Month 2 | 1 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 52 | 56 | 26
  LYM [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 51 | 53 | 24
  LYM [pre-vacc Normal; post-vacc Normal] Month 4 | 49 | 50 | 23
  LYM [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 51 | 53 | 24
  LYM [pre-vacc Normal; post-vacc Below] Month 4 | 2 | 3 | 0
  LYM [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 51 | 53 | 24
  LYM [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 0 | 1
  LYM [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 51 | 53 | 24
  LYM [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 51 | 53 | 24
  LYM [pre-vacc Normal; post-vacc Normal] Month 6 | 48 | 52 | 22
  LYM [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 51 | 53 | 24
  LYM [pre-vacc Normal; post-vacc Below] Month 6 | 3 | 1 | 0
  LYM [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 51 | 53 | 24
  LYM [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 2
  LYM [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 51 | 53 | 24
  LYM [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 50 | 52 | 23
  LYM [pre-vacc Normal; post-vacc Normal] Month 7 | 48 | 49 | 22
  LYM [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 50 | 52 | 23
  LYM [pre-vacc Normal; post-vacc Below] Month 7 | 2 | 3 | 0
  LYM [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 50 | 52 | 23
  LYM [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 0 | 1
  LYM [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 50 | 52 | 23
  LYM [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Normal] Day 7: number analyzed (Participants) | 2 | 1 | 1
  LYM [pre-vacc Low; post-vacc Normal] Day 7 | 2 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Day 7: number analyzed (Participants) | 2 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Day 7 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Above] Day 7: number analyzed (Participants) | 2 | 1 | 1
  LYM [pre-vacc Low; post-vacc Above] Day 7 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Missing] Day 7: number analyzed (Participants) | 2 | 1 | 1
  LYM [pre-vacc Low; post-vacc Missing] Day 7 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Normal] Month 1 | 3 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 1 | 2 | 0 | 0
  LYM [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Normal] Month 2 | 4 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 2 | 1 | 0 | 0
  LYM [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Normal] Month 4 | 3 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 4 | 2 | 0 | 0
  LYM [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Normal] Month 6 | 3 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 6 | 2 | 0 | 0
  LYM [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Normal] Month 7 | 3 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 7 | 2 | 0 | 0
  LYM [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Normal] Day 7: number analyzed (Participants) | 1 | 0 | 0
  LYM [pre-vacc High; post-vacc Normal] Day 7 | 1 | 0 | 0
  LYM [pre-vacc High; post-vacc Below] Day 7: number analyzed (Participants) | 1 | 0 | 0
  LYM [pre-vacc High; post-vacc Below] Day 7 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Above] Day 7: number analyzed (Participants) | 1 | 0 | 0
  LYM [pre-vacc High; post-vacc Above] Day 7 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Missing] Day 7: number analyzed (Participants) | 1 | 0 | 0
  LYM [pre-vacc High; post-vacc Missing] Day 7 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Normal] Month 1: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Normal] Month 1 | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 1: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 1 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Above] Month 1: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Above] Month 1 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Missing] Month 1: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Missing] Month 1 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Normal] Month 2: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Normal] Month 2 | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 2: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 2 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Above] Month 2: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Above] Month 2 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Missing] Month 2: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Missing] Month 2 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Normal] Month 4: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Normal] Month 4 | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 4: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 4 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Above] Month 4: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Above] Month 4 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Missing] Month 4: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Missing] Month 4 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Normal] Month 6: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Normal] Month 6 | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 6: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 6 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Above] Month 6: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Above] Month 6 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Missing] Month 6: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Missing] Month 6 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Normal] Month 7: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Normal] Month 7 | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 7: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 7 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Above] Month 7: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Above] Month 7 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Missing] Month 7: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Missing] Month 7 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 13 | 14 | 15
  MON [pre-vacc Normal; post-vacc Normal] Day 7 | 13 | 14 | 15
  MON [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 13 | 14 | 15
  MON [pre-vacc Normal; post-vacc Below] Day 7 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 13 | 14 | 15
  MON [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 13 | 14 | 15
  MON [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Normal] Month 1 | 56 | 54 | 28
  MON [pre-vacc Normal; post-vacc Below] Month 1 | 1 | 1 | 1
  MON [pre-vacc Normal; post-vacc Above] Month 1 | 0 | 1 | 0
  MON [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 55 | 56 | 28
  MON [pre-vacc Normal; post-vacc Normal] Month 2 | 52 | 55 | 28
  MON [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 55 | 56 | 28
  MON [pre-vacc Normal; post-vacc Below] Month 2 | 2 | 1 | 0
  MON [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 55 | 56 | 28
  MON [pre-vacc Normal; post-vacc Above] Month 2 | 1 | 0 | 0
  MON [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 55 | 56 | 28
  MON [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 54 | 53 | 26
  MON [pre-vacc Normal; post-vacc Normal] Month 4 | 51 | 52 | 26
  MON [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 54 | 53 | 26
  MON [pre-vacc Normal; post-vacc Below] Month 4 | 3 | 1 | 0
  MON [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 54 | 53 | 26
  MON [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 54 | 53 | 26
  MON [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 54 | 53 | 26
  MON [pre-vacc Normal; post-vacc Normal] Month 6 | 53 | 52 | 26
  MON [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 54 | 53 | 26
  MON [pre-vacc Normal; post-vacc Below] Month 6 | 1 | 1 | 0
  MON [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 54 | 53 | 26
  MON [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 54 | 53 | 26
  MON [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 53 | 52 | 25
  MON [pre-vacc Normal; post-vacc Normal] Month 7 | 50 | 50 | 24
  MON [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 53 | 52 | 25
  MON [pre-vacc Normal; post-vacc Below] Month 7 | 3 | 2 | 1
  MON [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 53 | 52 | 25
  MON [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 53 | 52 | 25
  MON [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Normal] Day 7: number analyzed (Participants) | 2 | 1 | 0
  MON [pre-vacc Low; post-vacc Normal] Day 7 | 2 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Day 7: number analyzed (Participants) | 2 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Day 7 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Above] Day 7: number analyzed (Participants) | 2 | 1 | 0
  MON [pre-vacc Low; post-vacc Above] Day 7 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Missing] Day 7: number analyzed (Participants) | 2 | 1 | 0
  MON [pre-vacc Low; post-vacc Missing] Day 7 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 1 | 2 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 1 | 1 | 0 | 0
  MON [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 2 | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 2 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 4 | 2 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 4 | 1 | 0 | 0
  MON [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 6 | 1 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 6 | 2 | 0 | 0
  MON [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 7 | 1 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 7 | 2 | 0 | 0
  MON [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0

13. Primary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Haemoglobin and Haematocrit Parameters at Day 7 and Months 1, 2, 4, 6 and 7
Description: Haematological laboratory parameters assessed were haemoglobin (Hgb) and haematocrit (Hct). For each parameter and by pre-vaccination status, it was assessed whether the post-vaccination values of the parameter were above, below or in the normal range (missing values are also indicated).
Time Frame: At Day 7 and Months 1, 2, 4, 6 and 7
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 49 | 48 | 26
Participants
  Hgb [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 14 | 14 | 13
  Hgb [pre-vacc Normal; post-vacc Normal] Day 7 | 13 | 11 | 13
  Hgb [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 14 | 14 | 13
  Hgb [pre-vacc Normal; post-vacc Below] Day 7 | 1 | 3 | 0
  Hgb [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 14 | 14 | 13
  Hgb [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 14 | 14 | 13
  Hgb [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Normal] Month 1: number analyzed (Participants) | 49 | 48 | 25
  Hgb [pre-vacc Normal; post-vacc Normal] Month 1 | 46 | 43 | 23
  Hgb [pre-vacc Normal; post-vacc Below] Month 1: number analyzed (Participants) | 49 | 48 | 25
  Hgb [pre-vacc Normal; post-vacc Below] Month 1 | 3 | 5 | 2
  Hgb [pre-vacc Normal; post-vacc Above] Month 1: number analyzed (Participants) | 49 | 48 | 25
  Hgb [pre-vacc Normal; post-vacc Above] Month 1 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Missing] Month 1: number analyzed (Participants) | 49 | 48 | 25
  Hgb [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 47 | 48 | 24
  Hgb [pre-vacc Normal; post-vacc Normal] Month 2 | 46 | 43 | 24
  Hgb [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 47 | 48 | 24
  Hgb [pre-vacc Normal; post-vacc Below] Month 2 | 1 | 4 | 0
  Hgb [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 47 | 48 | 24
  Hgb [pre-vacc Normal; post-vacc Above] Month 2 | 0 | 1 | 0
  Hgb [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 47 | 48 | 24
  Hgb [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 47 | 46 | 23
  Hgb [pre-vacc Normal; post-vacc Normal] Month 4 | 46 | 43 | 23
  Hgb [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 47 | 46 | 23
  Hgb [pre-vacc Normal; post-vacc Below] Month 4 | 1 | 3 | 0
  Hgb [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 47 | 46 | 23
  Hgb [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 47 | 46 | 23
  Hgb [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 47 | 45 | 23
  Hgb [pre-vacc Normal; post-vacc Normal] Month 6 | 42 | 39 | 23
  Hgb [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 47 | 45 | 23
  Hgb [pre-vacc Normal; post-vacc Below] Month 6 | 5 | 6 | 0
  Hgb [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 47 | 45 | 23
  Hgb [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 47 | 45 | 23
  Hgb [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 46 | 45 | 22
  Hgb [pre-vacc Normal; post-vacc Normal] Month 7 | 43 | 38 | 22
  Hgb [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 46 | 45 | 22
  Hgb [pre-vacc Normal; post-vacc Below] Month 7 | 3 | 7 | 0
  Hgb [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 46 | 45 | 22
  Hgb [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 46 | 45 | 22
  Hgb [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Normal] Day 7: number analyzed (Participants) | 1 | 1 | 2
  Hgb [pre-vacc Low; post-vacc Normal] Day 7 | 0 | 0 | 1
  Hgb [pre-vacc Low; post-vacc Below] Day 7: number analyzed (Participants) | 1 | 1 | 2
  Hgb [pre-vacc Low; post-vacc Below] Day 7 | 1 | 1 | 1
  Hgb [pre-vacc Low; post-vacc Above] Day 7: number analyzed (Participants) | 1 | 1 | 2
  Hgb [pre-vacc Low; post-vacc Above] Day 7 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Missing] Day 7: number analyzed (Participants) | 1 | 1 | 2
  Hgb [pre-vacc Low; post-vacc Missing] Day 7 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 11 | 9 | 4
  Hgb [pre-vacc Low; post-vacc Normal] Month 1 | 1 | 6 | 3
  Hgb [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 11 | 9 | 4
  Hgb [pre-vacc Low; post-vacc Below] Month 1 | 10 | 3 | 1
  Hgb [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 11 | 9 | 4
  Hgb [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 11 | 9 | 4
  Hgb [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 11 | 9 | 4
  Hgb [pre-vacc Low; post-vacc Normal] Month 2 | 3 | 2 | 3
  Hgb [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 11 | 9 | 4
  Hgb [pre-vacc Low; post-vacc Below] Month 2 | 8 | 7 | 1
  Hgb [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 11 | 9 | 4
  Hgb [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 11 | 9 | 4
  Hgb [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 10 | 8 | 3
  Hgb [pre-vacc Low; post-vacc Normal] Month 4 | 5 | 4 | 2
  Hgb [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 10 | 8 | 3
  Hgb [pre-vacc Low; post-vacc Below] Month 4 | 5 | 4 | 1
  Hgb [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 10 | 8 | 3
  Hgb [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 10 | 8 | 3
  Hgb [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 10 | 9 | 3
  Hgb [pre-vacc Low; post-vacc Normal] Month 6 | 6 | 3 | 2
  Hgb [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 10 | 9 | 3
  Hgb [pre-vacc Low; post-vacc Below] Month 6 | 4 | 6 | 1
  Hgb [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 10 | 9 | 3
  Hgb [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 10 | 9 | 3
  Hgb [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 10 | 8 | 3
  Hgb [pre-vacc Low; post-vacc Normal] Month 7 | 4 | 2 | 2
  Hgb [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 10 | 8 | 3
  Hgb [pre-vacc Low; post-vacc Below] Month 7 | 6 | 6 | 1
  Hgb [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 10 | 8 | 3
  Hgb [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 10 | 8 | 3
  Hgb [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 14 | 14 | 14
  Hct [pre-vacc Normal; post-vacc Normal] Day 7 | 11 | 11 | 13
  Hct [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 14 | 14 | 14
  Hct [pre-vacc Normal; post-vacc Below] Day 7 | 3 | 3 | 1
  Hct [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 14 | 14 | 14
  Hct [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 14 | 14 | 14
  Hct [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Normal] Month 1: number analyzed (Participants) | 44 | 43 | 26
  Hct [pre-vacc Normal; post-vacc Normal] Month 1 | 42 | 37 | 22
  Hct [pre-vacc Normal; post-vacc Below] Month 1: number analyzed (Participants) | 44 | 43 | 26
  Hct [pre-vacc Normal; post-vacc Below] Month 1 | 2 | 6 | 4
  Hct [pre-vacc Normal; post-vacc Above] Month 1: number analyzed (Participants) | 44 | 43 | 26
  Hct [pre-vacc Normal; post-vacc Above] Month 1 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Missing] Month 1: number analyzed (Participants) | 44 | 43 | 26
  Hct [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 42 | 43 | 25
  Hct [pre-vacc Normal; post-vacc Normal] Month 2 | 37 | 36 | 24
  Hct [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 42 | 43 | 25
  Hct [pre-vacc Normal; post-vacc Below] Month 2 | 5 | 6 | 1
  Hct [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 42 | 43 | 25
  Hct [pre-vacc Normal; post-vacc Above] Month 2 | 0 | 1 | 0
  Hct [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 42 | 43 | 25
  Hct [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 42 | 41 | 24
  Hct [pre-vacc Normal; post-vacc Normal] Month 4 | 38 | 36 | 24
  Hct [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 42 | 41 | 24
  Hct [pre-vacc Normal; post-vacc Below] Month 4 | 4 | 5 | 0
  Hct [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 42 | 41 | 24
  Hct [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 42 | 41 | 24
  Hct [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 42 | 40 | 24
  Hct [pre-vacc Normal; post-vacc Normal] Month 6 | 36 | 33 | 22
  Hct [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 42 | 40 | 24
  Hct [pre-vacc Normal; post-vacc Below] Month 6 | 6 | 7 | 1
  Hct [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 42 | 40 | 24
  Hct [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 1
  Hct [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 42 | 40 | 24
  Hct [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 41 | 40 | 23
  Hct [pre-vacc Normal; post-vacc Normal] Month 7 | 34 | 30 | 20
  Hct [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 41 | 40 | 23
  Hct [pre-vacc Normal; post-vacc Below] Month 7 | 7 | 10 | 2
  Hct [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 41 | 40 | 23
  Hct [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 0 | 1
  Hct [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 41 | 40 | 23
  Hct [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Normal] Day 7: number analyzed (Participants) | 1 | 1 | 1
  Hct [pre-vacc Low; post-vacc Normal] Day 7 | 0 | 0 | 1
  Hct [pre-vacc Low; post-vacc Below] Day 7: number analyzed (Participants) | 1 | 1 | 1
  Hct [pre-vacc Low; post-vacc Below] Day 7 | 1 | 1 | 0
  Hct [pre-vacc Low; post-vacc Above] Day 7: number analyzed (Participants) | 1 | 1 | 1
  Hct [pre-vacc Low; post-vacc Above] Day 7 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Missing] Day 7: number analyzed (Participants) | 1 | 1 | 1
  Hct [pre-vacc Low; post-vacc Missing] Day 7 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 16 | 13 | 3
  Hct [pre-vacc Low; post-vacc Normal] Month 1 | 4 | 2 | 1
  Hct [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 16 | 13 | 3
  Hct [pre-vacc Low; post-vacc Below] Month 1 | 12 | 11 | 2
  Hct [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 16 | 13 | 3
  Hct [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 16 | 13 | 3
  Hct [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 16 | 13 | 3
  Hct [pre-vacc Low; post-vacc Normal] Month 2 | 4 | 3 | 2
  Hct [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 16 | 13 | 3
  Hct [pre-vacc Low; post-vacc Below] Month 2 | 12 | 10 | 1
  Hct [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 16 | 13 | 3
  Hct [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 16 | 13 | 3
  Hct [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 15 | 12 | 2
  Hct [pre-vacc Low; post-vacc Normal] Month 4 | 6 | 3 | 1
  Hct [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 15 | 12 | 2
  Hct [pre-vacc Low; post-vacc Below] Month 4 | 9 | 9 | 1
  Hct [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 15 | 12 | 2
  Hct [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 15 | 12 | 2
  Hct [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 15 | 13 | 2
  Hct [pre-vacc Low; post-vacc Normal] Month 6 | 8 | 4 | 2
  Hct [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 15 | 13 | 2
  Hct [pre-vacc Low; post-vacc Below] Month 6 | 7 | 9 | 0
  Hct [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 15 | 13 | 2
  Hct [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 15 | 13 | 2
  Hct [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 15 | 12 | 2
  Hct [pre-vacc Low; post-vacc Normal] Month 7 | 8 | 3 | 2
  Hct [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 15 | 12 | 2
  Hct [pre-vacc Low; post-vacc Below] Month 7 | 7 | 9 | 0
  Hct [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 15 | 12 | 2
  Hct [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 15 | 12 | 2
  Hct [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 1: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 1 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Below] Month 1: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 1 | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 1: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 1 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 1: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 1 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 2: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 2 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Below] Month 2: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 2 | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 2: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 2 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 2: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 2 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 4: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 4 | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 4: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 4 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Above] Month 4: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 4 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 4: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 4 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 6: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 6 | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 6: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 6 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Above] Month 6: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 6 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 6: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 6 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 7: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 7 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Below] Month 7: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 7 | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 7: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 7 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 7: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 7 | 0 | 0 | 0

14. Primary Outcome: Number of Subjects With Clinically Relevant Abnormalities in Eosinophils, Basophils and Creatinine Parameters at Day 7 and Months 1, 2, 4, 6 and 7
Description: Haematological and biochemical laboratory parameters assessed were eosinophils (EOS), basophils (BAS) and creatinine (CREA). For each parameter and by pre-vaccination status, it was assessed whether the post-vaccination values of the parameter were above, below or in the normal range (missing values are also indicated).
Time Frame: At Day 7 and at Months 1, 2, 4, 6 and 7
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 60 | 57 | 29
Participants
  EOS [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 13 | 14 | 15
  EOS [pre-vacc Normal; post-vacc Normal] Day 7 | 13 | 13 | 15
  EOS [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 13 | 14 | 15
  EOS [pre-vacc Normal; post-vacc Below] Day 7 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 13 | 14 | 15
  EOS [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 1 | 0
  EOS [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 13 | 14 | 15
  EOS [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Normal] Month 1: number analyzed (Participants) | 54 | 54 | 28
  EOS [pre-vacc Normal; post-vacc Normal] Month 1 | 53 | 52 | 28
  EOS [pre-vacc Normal; post-vacc Below] Month 1: number analyzed (Participants) | 54 | 54 | 28
  EOS [pre-vacc Normal; post-vacc Below] Month 1 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Above] Month 1: number analyzed (Participants) | 54 | 54 | 28
  EOS [pre-vacc Normal; post-vacc Above] Month 1 | 1 | 2 | 0
  EOS [pre-vacc Normal; post-vacc Missing] Month 1: number analyzed (Participants) | 54 | 54 | 28
  EOS [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 52 | 54 | 27
  EOS [pre-vacc Normal; post-vacc Normal] Month 2 | 51 | 51 | 26
  EOS [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 52 | 54 | 27
  EOS [pre-vacc Normal; post-vacc Below] Month 2 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 52 | 54 | 27
  EOS [pre-vacc Normal; post-vacc Above] Month 2 | 1 | 3 | 1
  EOS [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 52 | 54 | 27
  EOS [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 51 | 51 | 25
  EOS [pre-vacc Normal; post-vacc Normal] Month 4 | 48 | 49 | 25
  EOS [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 51 | 51 | 25
  EOS [pre-vacc Normal; post-vacc Below] Month 4 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 51 | 51 | 25
  EOS [pre-vacc Normal; post-vacc Above] Month 4 | 3 | 2 | 0
  EOS [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 51 | 51 | 25
  EOS [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 51 | 51 | 25
  EOS [pre-vacc Normal; post-vacc Normal] Month 6 | 50 | 51 | 25
  EOS [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 51 | 51 | 25
  EOS [pre-vacc Normal; post-vacc Below] Month 6 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 51 | 51 | 25
  EOS [pre-vacc Normal; post-vacc Above] Month 6 | 1 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 51 | 51 | 25
  EOS [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 50 | 50 | 24
  EOS [pre-vacc Normal; post-vacc Normal] Month 7 | 50 | 49 | 24
  EOS [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 50 | 50 | 24
  EOS [pre-vacc Normal; post-vacc Below] Month 7 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 50 | 50 | 24
  EOS [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 1 | 0
  EOS [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 50 | 50 | 24
  EOS [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Normal] Day 7: number analyzed (Participants) | 2 | 1 | 0
  EOS [pre-vacc High; post-vacc Normal] Day 7 | 1 | 1 | 0
  EOS [pre-vacc High; post-vacc Below] Day 7: number analyzed (Participants) | 2 | 1 | 0
  EOS [pre-vacc High; post-vacc Below] Day 7 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Above] Day 7: number analyzed (Participants) | 2 | 1 | 0
  EOS [pre-vacc High; post-vacc Above] Day 7 | 1 | 0 | 0
  EOS [pre-vacc High; post-vacc Missing] Day 7: number analyzed (Participants) | 2 | 1 | 0
  EOS [pre-vacc High; post-vacc Missing] Day 7 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Normal] Month 1: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Normal] Month 1 | 5 | 2 | 1
  EOS [pre-vacc High; post-vacc Below] Month 1: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Below] Month 1 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Above] Month 1: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Above] Month 1 | 1 | 1 | 0
  EOS [pre-vacc High; post-vacc Missing] Month 1: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Missing] Month 1 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Normal] Month 2: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Normal] Month 2 | 3 | 2 | 1
  EOS [pre-vacc High; post-vacc Below] Month 2: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Below] Month 2 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Above] Month 2: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Above] Month 2 | 3 | 1 | 0
  EOS [pre-vacc High; post-vacc Missing] Month 2: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Missing] Month 2 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Normal] Month 4: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Normal] Month 4 | 5 | 1 | 1
  EOS [pre-vacc High; post-vacc Below] Month 4: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Below] Month 4 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Above] Month 4: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Above] Month 4 | 1 | 2 | 0
  EOS [pre-vacc High; post-vacc Missing] Month 4: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Missing] Month 4 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Normal] Month 6: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Normal] Month 6 | 4 | 2 | 0
  EOS [pre-vacc High; post-vacc Below] Month 6: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Below] Month 6 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Above] Month 6: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Above] Month 6 | 2 | 1 | 1
  EOS [pre-vacc High; post-vacc Missing] Month 6: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Missing] Month 6 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Normal] Month 7: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Normal] Month 7 | 4 | 1 | 0
  EOS [pre-vacc High; post-vacc Below] Month 7: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Below] Month 7 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Above] Month 7: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Above] Month 7 | 2 | 2 | 1
  EOS [pre-vacc High; post-vacc Missing] Month 7: number analyzed (Participants) | 6 | 3 | 1
  EOS [pre-vacc High; post-vacc Missing] Month 7 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 15 | 15 | 15
  BAS [pre-vacc Normal; post-vacc Normal] Day 7 | 15 | 15 | 15
  BAS [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 15 | 15 | 15
  BAS [pre-vacc Normal; post-vacc Below] Day 7 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 15 | 15 | 15
  BAS [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 15 | 15 | 15
  BAS [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Normal] Month 1 | 60 | 57 | 29
  BAS [pre-vacc Normal; post-vacc Below] Month 1 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Above] Month 1 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 58 | 57 | 28
  BAS [pre-vacc Normal; post-vacc Normal] Month 2 | 58 | 57 | 28
  BAS [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 58 | 57 | 28
  BAS [pre-vacc Normal; post-vacc Below] Month 2 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 58 | 57 | 28
  BAS [pre-vacc Normal; post-vacc Above] Month 2 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 58 | 57 | 28
  BAS [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Normal] Month 4 | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Below] Month 4 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Normal] Month 6 | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Below] Month 6 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 57 | 54 | 26
  BAS [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 56 | 53 | 25
  BAS [pre-vacc Normal; post-vacc Normal] Month 7 | 56 | 53 | 25
  BAS [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 56 | 53 | 25
  BAS [pre-vacc Normal; post-vacc Below] Month 7 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 56 | 53 | 25
  BAS [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 56 | 53 | 25
  BAS [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 7 | 7 | 12
  CREA [pre-vacc Normal; post-vacc Normal] Day 7 | 6 | 4 | 11
  CREA [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 7 | 7 | 12
  CREA [pre-vacc Normal; post-vacc Below] Day 7 | 1 | 3 | 1
  CREA [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 7 | 7 | 12
  CREA [pre-vacc Normal; post-vacc Above] Day 7 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 7 | 7 | 12
  CREA [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Normal] Month 1: number analyzed (Participants) | 28 | 37 | 22
  CREA [pre-vacc Normal; post-vacc Normal] Month 1 | 24 | 29 | 17
  CREA [pre-vacc Normal; post-vacc Below] Month 1: number analyzed (Participants) | 28 | 37 | 22
  CREA [pre-vacc Normal; post-vacc Below] Month 1 | 4 | 8 | 5
  CREA [pre-vacc Normal; post-vacc Above] Month 1: number analyzed (Participants) | 28 | 37 | 22
  CREA [pre-vacc Normal; post-vacc Above] Month 1 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Missing] Month 1: number analyzed (Participants) | 28 | 37 | 22
  CREA [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 27 | 37 | 21
  CREA [pre-vacc Normal; post-vacc Normal] Month 2 | 26 | 30 | 15
  CREA [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 27 | 37 | 21
  CREA [pre-vacc Normal; post-vacc Below] Month 2 | 1 | 7 | 6
  CREA [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 27 | 37 | 21
  CREA [pre-vacc Normal; post-vacc Above] Month 2 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 27 | 37 | 21
  CREA [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 26 | 35 | 20
  CREA [pre-vacc Normal; post-vacc Normal] Month 4 | 24 | 26 | 17
  CREA [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 26 | 35 | 20
  CREA [pre-vacc Normal; post-vacc Below] Month 4 | 2 | 9 | 3
  CREA [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 26 | 35 | 20
  CREA [pre-vacc Normal; post-vacc Above] Month 4 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 26 | 35 | 20
  CREA [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 26 | 34 | 20
  CREA [pre-vacc Normal; post-vacc Normal] Month 6 | 20 | 22 | 17
  CREA [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 26 | 34 | 20
  CREA [pre-vacc Normal; post-vacc Below] Month 6 | 6 | 12 | 3
  CREA [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 26 | 34 | 20
  CREA [pre-vacc Normal; post-vacc Above] Month 6 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 26 | 34 | 20
  CREA [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 25 | 35 | 20
  CREA [pre-vacc Normal; post-vacc Normal] Month 7 | 22 | 24 | 15
  CREA [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 25 | 35 | 20
  CREA [pre-vacc Normal; post-vacc Below] Month 7 | 3 | 11 | 5
  CREA [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 25 | 35 | 20
  CREA [pre-vacc Normal; post-vacc Above] Month 7 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 25 | 35 | 20
  CREA [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Normal] Day 7: number analyzed (Participants) | 8 | 8 | 3
  CREA [pre-vacc Low; post-vacc Normal] Day 7 | 2 | 2 | 0
  CREA [pre-vacc Low; post-vacc Below] Day 7: number analyzed (Participants) | 8 | 8 | 3
  CREA [pre-vacc Low; post-vacc Below] Day 7 | 6 | 6 | 3
  CREA [pre-vacc Low; post-vacc Above] Day 7: number analyzed (Participants) | 8 | 8 | 3
  CREA [pre-vacc Low; post-vacc Above] Day 7 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Missing] Day 7: number analyzed (Participants) | 8 | 8 | 3
  CREA [pre-vacc Low; post-vacc Missing] Day 7 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 32 | 20 | 7
  CREA [pre-vacc Low; post-vacc Normal] Month 1 | 5 | 7 | 1
  CREA [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 32 | 20 | 7
  CREA [pre-vacc Low; post-vacc Below] Month 1 | 27 | 13 | 6
  CREA [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 32 | 20 | 7
  CREA [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 32 | 20 | 7
  CREA [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 31 | 20 | 7
  CREA [pre-vacc Low; post-vacc Normal] Month 2 | 8 | 5 | 2
  CREA [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 31 | 20 | 7
  CREA [pre-vacc Low; post-vacc Below] Month 2 | 23 | 15 | 5
  CREA [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 31 | 20 | 7
  CREA [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 31 | 20 | 7
  CREA [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 31 | 19 | 6
  CREA [pre-vacc Low; post-vacc Normal] Month 4 | 6 | 7 | 1
  CREA [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 31 | 19 | 6
  CREA [pre-vacc Low; post-vacc Below] Month 4 | 25 | 12 | 5
  CREA [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 31 | 19 | 6
  CREA [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 31 | 19 | 6
  CREA [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 31 | 20 | 6
  CREA [pre-vacc Low; post-vacc Normal] Month 6 | 10 | 7 | 3
  CREA [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 31 | 20 | 6
  CREA [pre-vacc Low; post-vacc Below] Month 6 | 21 | 13 | 3
  CREA [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 31 | 20 | 6
  CREA [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 31 | 20 | 6
  CREA [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 31 | 18 | 5
  CREA [pre-vacc Low; post-vacc Normal] Month 7 | 7 | 5 | 1
  CREA [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 31 | 18 | 5
  CREA [pre-vacc Low; post-vacc Below] Month 7 | 24 | 13 | 4
  CREA [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 31 | 18 | 5
  CREA [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 31 | 18 | 5
  CREA [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0

15. Primary Outcome: Number of Subjects With Clinically Relevant Abnormalities in Alanine Aminotransferase Parameter at Day 7 and Months 1, 2, 4, 6 and 7
Description: Biochemical laboratory parameter assessed was alanine aminotransferase (ALAT). By pre-vaccination status, it was assessed whether the post-vaccination values of the parameter were above, below or in the normal range (missing values are also indicated).
Time Frame: At Day 7 and Months 1, 2, 4, 6 and 7
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 50 | 46 | 26
Participants
  ALAT [pre-vacc Normal; post-vacc Normal] Day 7: number analyzed (Participants) | 11 | 12 | 12
  ALAT [pre-vacc Normal; post-vacc Normal] Day 7 | 10 | 12 | 12
  ALAT [pre-vacc Normal; post-vacc Below] Day 7: number analyzed (Participants) | 11 | 12 | 12
  ALAT [pre-vacc Normal; post-vacc Below] Day 7 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Above] Day 7: number analyzed (Participants) | 11 | 12 | 12
  ALAT [pre-vacc Normal; post-vacc Above] Day 7 | 1 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Missing] Day 7: number analyzed (Participants) | 11 | 12 | 12
  ALAT [pre-vacc Normal; post-vacc Missing] Day 7 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Normal] Month 1 | 48 | 45 | 25
  ALAT [pre-vacc Normal; post-vacc Below] Month 1 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Above] Month 1 | 2 | 1 | 1
  ALAT [pre-vacc Normal; post-vacc Missing] Month 1 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Normal] Month 2: number analyzed (Participants) | 48 | 46 | 25
  ALAT [pre-vacc Normal; post-vacc Normal] Month 2 | 47 | 40 | 24
  ALAT [pre-vacc Normal; post-vacc Below] Month 2: number analyzed (Participants) | 48 | 46 | 25
  ALAT [pre-vacc Normal; post-vacc Below] Month 2 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Above] Month 2: number analyzed (Participants) | 48 | 46 | 25
  ALAT [pre-vacc Normal; post-vacc Above] Month 2 | 1 | 6 | 1
  ALAT [pre-vacc Normal; post-vacc Missing] Month 2: number analyzed (Participants) | 48 | 46 | 25
  ALAT [pre-vacc Normal; post-vacc Missing] Month 2 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Normal] Month 4: number analyzed (Participants) | 47 | 45 | 23
  ALAT [pre-vacc Normal; post-vacc Normal] Month 4 | 44 | 42 | 23
  ALAT [pre-vacc Normal; post-vacc Below] Month 4: number analyzed (Participants) | 47 | 45 | 23
  ALAT [pre-vacc Normal; post-vacc Below] Month 4 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Above] Month 4: number analyzed (Participants) | 47 | 45 | 23
  ALAT [pre-vacc Normal; post-vacc Above] Month 4 | 3 | 3 | 0
  ALAT [pre-vacc Normal; post-vacc Missing] Month 4: number analyzed (Participants) | 47 | 45 | 23
  ALAT [pre-vacc Normal; post-vacc Missing] Month 4 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Normal] Month 6: number analyzed (Participants) | 47 | 45 | 23
  ALAT [pre-vacc Normal; post-vacc Normal] Month 6 | 46 | 41 | 21
  ALAT [pre-vacc Normal; post-vacc Below] Month 6: number analyzed (Participants) | 47 | 45 | 23
  ALAT [pre-vacc Normal; post-vacc Below] Month 6 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Above] Month 6: number analyzed (Participants) | 47 | 45 | 23
  ALAT [pre-vacc Normal; post-vacc Above] Month 6 | 1 | 4 | 2
  ALAT [pre-vacc Normal; post-vacc Missing] Month 6: number analyzed (Participants) | 47 | 45 | 23
  ALAT [pre-vacc Normal; post-vacc Missing] Month 6 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Normal] Month 7: number analyzed (Participants) | 46 | 45 | 22
  ALAT [pre-vacc Normal; post-vacc Normal] Month 7 | 40 | 40 | 22
  ALAT [pre-vacc Normal; post-vacc Below] Month 7: number analyzed (Participants) | 46 | 45 | 22
  ALAT [pre-vacc Normal; post-vacc Below] Month 7 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Above] Month 7: number analyzed (Participants) | 46 | 45 | 22
  ALAT [pre-vacc Normal; post-vacc Above] Month 7 | 6 | 5 | 0
  ALAT [pre-vacc Normal; post-vacc Missing] Month 7: number analyzed (Participants) | 46 | 45 | 22
  ALAT [pre-vacc Normal; post-vacc Missing] Month 7 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 1: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 1 | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 1: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 1 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 1: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 1 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 1: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 1 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 2: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 2 | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 2: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 2 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 2: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 2 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 2: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 2 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 4: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 4 | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 4: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 4 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 4: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 4 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 4: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 4 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 6: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 6 | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 6: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 6 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 6: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 6 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 6: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 6 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 7: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 7 | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 7: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 7 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 7: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 7 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 7: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 7 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Normal] Day 7: number analyzed (Participants) | 4 | 3 | 3
  ALAT [pre-vacc High; post-vacc Normal] Day 7 | 2 | 2 | 2
  ALAT [pre-vacc High; post-vacc Below] Day 7: number analyzed (Participants) | 4 | 3 | 3
  ALAT [pre-vacc High; post-vacc Below] Day 7 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Above] Day 7: number analyzed (Participants) | 4 | 3 | 3
  ALAT [pre-vacc High; post-vacc Above] Day 7 | 2 | 1 | 1
  ALAT [pre-vacc High; post-vacc Missing] Day 7: number analyzed (Participants) | 4 | 3 | 3
  ALAT [pre-vacc High; post-vacc Missing] Day 7 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Normal] Month 1: number analyzed (Participants) | 9 | 11 | 3
  ALAT [pre-vacc High; post-vacc Normal] Month 1 | 6 | 6 | 2
  ALAT [pre-vacc High; post-vacc Below] Month 1: number analyzed (Participants) | 9 | 11 | 3
  ALAT [pre-vacc High; post-vacc Below] Month 1 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Above] Month 1: number analyzed (Participants) | 9 | 11 | 3
  ALAT [pre-vacc High; post-vacc Above] Month 1 | 3 | 5 | 1
  ALAT [pre-vacc High; post-vacc Missing] Month 1: number analyzed (Participants) | 9 | 11 | 3
  ALAT [pre-vacc High; post-vacc Missing] Month 1 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Normal] Month 2: number analyzed (Participants) | 9 | 11 | 3
  ALAT [pre-vacc High; post-vacc Normal] Month 2 | 9 | 8 | 1
  ALAT [pre-vacc High; post-vacc Below] Month 2: number analyzed (Participants) | 9 | 11 | 3
  ALAT [pre-vacc High; post-vacc Below] Month 2 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Above] Month 2: number analyzed (Participants) | 9 | 11 | 3
  ALAT [pre-vacc High; post-vacc Above] Month 2 | 0 | 3 | 2
  ALAT [pre-vacc High; post-vacc Missing] Month 2: number analyzed (Participants) | 9 | 11 | 3
  ALAT [pre-vacc High; post-vacc Missing] Month 2 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Normal] Month 4: number analyzed (Participants) | 9 | 9 | 3
  ALAT [pre-vacc High; post-vacc Normal] Month 4 | 9 | 7 | 1
  ALAT [pre-vacc High; post-vacc Below] Month 4: number analyzed (Participants) | 9 | 9 | 3
  ALAT [pre-vacc High; post-vacc Below] Month 4 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Above] Month 4: number analyzed (Participants) | 9 | 9 | 3
  ALAT [pre-vacc High; post-vacc Above] Month 4 | 0 | 2 | 2
  ALAT [pre-vacc High; post-vacc Missing] Month 4: number analyzed (Participants) | 9 | 9 | 3
  ALAT [pre-vacc High; post-vacc Missing] Month 4 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Normal] Month 6: number analyzed (Participants) | 9 | 9 | 3
  ALAT [pre-vacc High; post-vacc Normal] Month 6 | 7 | 6 | 2
  ALAT [pre-vacc High; post-vacc Below] Month 6: number analyzed (Participants) | 9 | 9 | 3
  ALAT [pre-vacc High; post-vacc Below] Month 6 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Above] Month 6: number analyzed (Participants) | 9 | 9 | 3
  ALAT [pre-vacc High; post-vacc Above] Month 6 | 2 | 3 | 1
  ALAT [pre-vacc High; post-vacc Missing] Month 6: number analyzed (Participants) | 9 | 9 | 3
  ALAT [pre-vacc High; post-vacc Missing] Month 6 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Normal] Month 7: number analyzed (Participants) | 9 | 8 | 3
  ALAT [pre-vacc High; post-vacc Normal] Month 7 | 7 | 5 | 2
  ALAT [pre-vacc High; post-vacc Below] Month 7: number analyzed (Participants) | 9 | 8 | 3
  ALAT [pre-vacc High; post-vacc Below] Month 7 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Above] Month 7: number analyzed (Participants) | 9 | 8 | 3
  ALAT [pre-vacc High; post-vacc Above] Month 7 | 2 | 3 | 1
  ALAT [pre-vacc High; post-vacc Missing] Month 7: number analyzed (Participants) | 9 | 8 | 3
  ALAT [pre-vacc High; post-vacc Missing] Month 7 | 0 | 0 | 0

16. Primary Outcome: Number of Subjects Reporting Clinically Relevant Abnormalities in Neutrophils, Platelets, Red Blood Cells and White Blood Cells at Month 10 and Month 12
Description: Haematological laboratory parameters assessed were neutrophils (NEU), platelets (PLA), red blood cells (RBC) and white blood cells (WBC). For each parameter and by pre-vaccination status, it was assessed whether the post-vaccination values of the parameter were above, below or in the normal range (missing values are also indicated).
Time Frame: At Month 10 and Month 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 51 | 50 | 24
Participants
  NEU [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 43 | 36 | 21
  NEU [pre-vacc Normal; post-vacc Normal] Month 10 | 32 | 30 | 16
  NEU [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 43 | 36 | 21
  NEU [pre-vacc Normal; post-vacc Below] Month 10 | 11 | 4 | 5
  NEU [pre-vacc Normal; post-vacc Above] Month 10: number analyzed (Participants) | 43 | 36 | 21
  NEU [pre-vacc Normal; post-vacc Above] Month 10 | 0 | 2 | 0
  NEU [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 43 | 36 | 21
  NEU [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 42 | 38 | 21
  NEU [pre-vacc Normal; post-vacc Normal] Month 12 | 29 | 32 | 17
  NEU [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 42 | 38 | 21
  NEU [pre-vacc Normal; post-vacc Below] Month 12 | 13 | 6 | 4
  NEU [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 42 | 38 | 21
  NEU [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 0 | 0
  NEU [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 42 | 38 | 21
  NEU [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Normal] Month 10 | 6 | 4 | 0
  NEU [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Below] Month 10 | 6 | 10 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 10: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 10 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Normal] Month 12 | 3 | 3 | 1
  NEU [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Below] Month 12 | 9 | 11 | 2
  NEU [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  NEU [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 12 | 14 | 3
  NEU [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 51 | 48 | 24
  PLA [pre-vacc Normal; post-vacc Normal] Month 10 | 48 | 47 | 24
  PLA [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 51 | 48 | 24
  PLA [pre-vacc Normal; post-vacc Below] Month 10 | 1 | 1 | 0
  PLA [pre-vacc Normal; post-vacc Above] Month 10: number analyzed (Participants) | 51 | 48 | 24
  PLA [pre-vacc Normal; post-vacc Above] Month 10 | 1 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 51 | 48 | 24
  PLA [pre-vacc Normal; post-vacc Missing] Month 10 | 1 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 50 | 50 | 24
  PLA [pre-vacc Normal; post-vacc Normal] Month 12 | 50 | 49 | 24
  PLA [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 50 | 50 | 24
  PLA [pre-vacc Normal; post-vacc Below] Month 12 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 50 | 50 | 24
  PLA [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 0 | 0
  PLA [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 50 | 50 | 24
  PLA [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 1 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 10 | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 10 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 10: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 10 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Normal] Month 12 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Below] Month 12 | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 1 | 0 | 0
  PLA [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 10: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 10 | 2 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 10: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 10 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Above] Month 10: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Above] Month 10 | 1 | 0 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 10: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 10 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 12: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Normal] Month 12 | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 12: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Below] Month 12 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Above] Month 12: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Above] Month 12 | 0 | 0 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 12: number analyzed (Participants) | 3 | 2 | 0
  PLA [pre-vacc High; post-vacc Missing] Month 12 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 48 | 43 | 24
  RBC [pre-vacc Normal; post-vacc Normal] Month 10 | 40 | 34 | 23
  RBC [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 48 | 43 | 24
  RBC [pre-vacc Normal; post-vacc Below] Month 10 | 8 | 9 | 1
  RBC [pre-vacc Normal; post-vacc Above] Month 10: number analyzed (Participants) | 48 | 43 | 24
  RBC [pre-vacc Normal; post-vacc Above] Month 10 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 48 | 43 | 24
  RBC [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 47 | 45 | 24
  RBC [pre-vacc Normal; post-vacc Normal] Month 12 | 40 | 40 | 24
  RBC [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 47 | 45 | 24
  RBC [pre-vacc Normal; post-vacc Below] Month 12 | 7 | 5 | 0
  RBC [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 47 | 45 | 24
  RBC [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 0 | 0
  RBC [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 47 | 45 | 24
  RBC [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 7 | 7 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 10 | 1 | 1 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 7 | 7 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 10 | 6 | 6 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 10: number analyzed (Participants) | 7 | 7 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 10 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 7 | 7 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 7 | 7 | 0
  RBC [pre-vacc Low; post-vacc Normal] Month 12 | 0 | 2 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 7 | 7 | 0
  RBC [pre-vacc Low; post-vacc Below] Month 12 | 7 | 5 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 7 | 7 | 0
  RBC [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 7 | 7 | 0
  RBC [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 42 | 43 | 22
  WBC [pre-vacc Normal; post-vacc Normal] Month 10 | 35 | 36 | 19
  WBC [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 42 | 43 | 22
  WBC [pre-vacc Normal; post-vacc Below] Month 10 | 7 | 6 | 3
  WBC [pre-vacc Normal; post-vacc Above] Month 10: number analyzed (Participants) | 42 | 43 | 22
  WBC [pre-vacc Normal; post-vacc Above] Month 10 | 0 | 1 | 0
  WBC [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 42 | 43 | 22
  WBC [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 41 | 45 | 22
  WBC [pre-vacc Normal; post-vacc Normal] Month 12 | 34 | 35 | 17
  WBC [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 41 | 45 | 22
  WBC [pre-vacc Normal; post-vacc Below] Month 12 | 7 | 10 | 5
  WBC [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 41 | 45 | 22
  WBC [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 0 | 0
  WBC [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 41 | 45 | 22
  WBC [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 13 | 7 | 2
  WBC [pre-vacc Low; post-vacc Normal] Month 10 | 6 | 4 | 1
  WBC [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 13 | 7 | 2
  WBC [pre-vacc Low; post-vacc Below] Month 10 | 7 | 3 | 1
  WBC [pre-vacc Low; post-vacc Above] Month 10: number analyzed (Participants) | 13 | 7 | 2
  WBC [pre-vacc Low; post-vacc Above] Month 10 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 13 | 7 | 2
  WBC [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 13 | 7 | 2
  WBC [pre-vacc Low; post-vacc Normal] Month 12 | 6 | 4 | 0
  WBC [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 13 | 7 | 2
  WBC [pre-vacc Low; post-vacc Below] Month 12 | 7 | 3 | 2
  WBC [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 13 | 7 | 2
  WBC [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  WBC [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 13 | 7 | 2
  WBC [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0

17. Primary Outcome: Number of Subjects With Clinically Relevant Abnormalities in Alanine Aminotransferase, Basophils, Creatinine, Eosinophils, Haematocrit, Haemoglobin, Lymphocytes and Monocytes Parameters at Month 10 and Month 12
Description: Haematological and biochemical laboratory parameters assessed were alanine aminotransferase (ALAT), basophils (BAS), creatinine (CREA), eosinophils (EOS), haematocrit (Hct), haemoglobin (Hgb), lymphocytes (LYM) and monocytes (MON). For each parameter and by pre-vaccination status, it was assessed whether the post-vaccination values of the parameter were above, below or in the normal range (missing values are also indicated).
Time Frame: At Month 10 and Month 12
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 55 | 52 | 24
Participants
  ALAT [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 45 | 44 | 21
  ALAT [pre-vacc Normal; post-vacc Normal] Month 10 | 44 | 40 | 20
  ALAT [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 45 | 44 | 21
  ALAT [pre-vacc Normal; post-vacc Below] Month 10 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Above] Month 10: number analyzed (Participants) | 45 | 44 | 21
  ALAT [pre-vacc Normal; post-vacc Above] Month 10 | 1 | 4 | 1
  ALAT [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 45 | 44 | 21
  ALAT [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 44 | 45 | 21
  ALAT [pre-vacc Normal; post-vacc Normal] Month 12 | 38 | 39 | 20
  ALAT [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 44 | 45 | 21
  ALAT [pre-vacc Normal; post-vacc Below] Month 12 | 0 | 0 | 0
  ALAT [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 44 | 45 | 21
  ALAT [pre-vacc Normal; post-vacc Above] Month 12 | 6 | 6 | 1
  ALAT [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 44 | 45 | 21
  ALAT [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 10 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 10 | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 10: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 10 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Normal] Month 12 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Below] Month 12 | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 1 | 0 | 0
  ALAT [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Normal] Month 10: number analyzed (Participants) | 9 | 6 | 3
  ALAT [pre-vacc High; post-vacc Normal] Month 10 | 8 | 4 | 1
  ALAT [pre-vacc High; post-vacc Below] Month 10: number analyzed (Participants) | 9 | 6 | 3
  ALAT [pre-vacc High; post-vacc Below] Month 10 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Above] Month 10: number analyzed (Participants) | 9 | 6 | 3
  ALAT [pre-vacc High; post-vacc Above] Month 10 | 1 | 2 | 2
  ALAT [pre-vacc High; post-vacc Missing] Month 10: number analyzed (Participants) | 9 | 6 | 3
  ALAT [pre-vacc High; post-vacc Missing] Month 10 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Normal] Month 12: number analyzed (Participants) | 9 | 7 | 3
  ALAT [pre-vacc High; post-vacc Normal] Month 12 | 8 | 5 | 2
  ALAT [pre-vacc High; post-vacc Below] Month 12: number analyzed (Participants) | 9 | 7 | 3
  ALAT [pre-vacc High; post-vacc Below] Month 12 | 0 | 0 | 0
  ALAT [pre-vacc High; post-vacc Above] Month 12: number analyzed (Participants) | 9 | 7 | 3
  ALAT [pre-vacc High; post-vacc Above] Month 12 | 1 | 2 | 1
  ALAT [pre-vacc High; post-vacc Missing] Month 12: number analyzed (Participants) | 9 | 7 | 3
  ALAT [pre-vacc High; post-vacc Missing] Month 12 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 55 | 50 | 24
  BAS [pre-vacc Normal; post-vacc Normal] Month 10 | 55 | 50 | 24
  BAS [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 55 | 50 | 24
  BAS [pre-vacc Normal; post-vacc Below] Month 10 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Above] Month 10: number analyzed (Participants) | 55 | 50 | 24
  BAS [pre-vacc Normal; post-vacc Above] Month 10 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 55 | 50 | 24
  BAS [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 54 | 52 | 24
  BAS [pre-vacc Normal; post-vacc Normal] Month 12 | 54 | 52 | 24
  BAS [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 54 | 52 | 24
  BAS [pre-vacc Normal; post-vacc Below] Month 12 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 54 | 52 | 24
  BAS [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 0 | 0
  BAS [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 54 | 52 | 24
  BAS [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 24 | 33 | 19
  CREA [pre-vacc Normal; post-vacc Normal] Month 10 | 20 | 22 | 15
  CREA [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 24 | 33 | 19
  CREA [pre-vacc Normal; post-vacc Below] Month 10 | 4 | 11 | 4
  CREA [pre-vacc Normal; post-vacc Above] Month 10: number analyzed (Participants) | 24 | 33 | 19
  CREA [pre-vacc Normal; post-vacc Above] Month 10 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 24 | 33 | 19
  CREA [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 24 | 34 | 19
  CREA [pre-vacc Normal; post-vacc Normal] Month 12 | 18 | 24 | 13
  CREA [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 24 | 34 | 19
  CREA [pre-vacc Normal; post-vacc Below] Month 12 | 6 | 10 | 6
  CREA [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 24 | 34 | 19
  CREA [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 0 | 0
  CREA [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 24 | 34 | 19
  CREA [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 31 | 17 | 5
  CREA [pre-vacc Low; post-vacc Normal] Month 10 | 11 | 4 | 2
  CREA [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 31 | 17 | 5
  CREA [pre-vacc Low; post-vacc Below] Month 10 | 20 | 13 | 3
  CREA [pre-vacc Low ; post-vacc Above] Month 10: number analyzed (Participants) | 31 | 17 | 5
  CREA [pre-vacc Low ; post-vacc Above] Month 10 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 31 | 17 | 5
  CREA [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 30 | 18 | 5
  CREA [pre-vacc Low; post-vacc Normal] Month 12 | 4 | 4 | 3
  CREA [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 30 | 18 | 5
  CREA [pre-vacc Low; post-vacc Below] Month 12 | 26 | 14 | 2
  CREA [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 30 | 18 | 5
  CREA [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  CREA [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 30 | 18 | 5
  CREA [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 49 | 48 | 24
  EOS [pre-vacc Normal; post-vacc Normal] Month 10 | 46 | 46 | 22
  EOS [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 49 | 48 | 24
  EOS [pre-vacc Normal; post-vacc Below] Month 10 | 0 | 0 | 0
  EOS [pre-vacc Normal ; post-vacc Above] Month 10: number analyzed (Participants) | 49 | 48 | 24
  EOS [pre-vacc Normal ; post-vacc Above] Month 10 | 3 | 2 | 2
  EOS [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 49 | 48 | 24
  EOS [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 48 | 50 | 24
  EOS [pre-vacc Normal; post-vacc Normal] Month 12 | 46 | 49 | 24
  EOS [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 48 | 50 | 24
  EOS [pre-vacc Normal; post-vacc Below] Month 12 | 0 | 0 | 0
  EOS [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 48 | 50 | 24
  EOS [pre-vacc Normal; post-vacc Above] Month 12 | 2 | 1 | 0
  EOS [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 48 | 50 | 24
  EOS [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Normal] Month 10: number analyzed (Participants) | 6 | 2 | 0
  EOS [pre-vacc High; post-vacc Normal] Month 10 | 3 | 2 | 0
  EOS [pre-vacc High; post-vacc Below] Month 10: number analyzed (Participants) | 6 | 2 | 0
  EOS [pre-vacc High; post-vacc Below] Month 10 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Above] Month 10: number analyzed (Participants) | 6 | 2 | 0
  EOS [pre-vacc High; post-vacc Above] Month 10 | 3 | 0 | 0
  EOS [pre-vacc High; post-vacc Missing] Month 10: number analyzed (Participants) | 6 | 2 | 0
  EOS [pre-vacc High; post-vacc Missing] Month 10 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Normal] Month 12: number analyzed (Participants) | 6 | 2 | 0
  EOS [pre-vacc High; post-vacc Normal] Month 12 | 4 | 2 | 0
  EOS [pre-vacc High; post-vacc Below] Month 12: number analyzed (Participants) | 6 | 2 | 0
  EOS [pre-vacc High; post-vacc Below] Month 12 | 0 | 0 | 0
  EOS [pre-vacc High; post-vacc Above] Month 12: number analyzed (Participants) | 6 | 2 | 0
  EOS [pre-vacc High; post-vacc Above] Month 12 | 2 | 0 | 0
  EOS [pre-vacc High; post-vacc Missing] Month 12: number analyzed (Participants) | 6 | 2 | 0
  EOS [pre-vacc High; post-vacc Missing] Month 12 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 41 | 38 | 22
  Hct [pre-vacc Normal; post-vacc Normal] Month 10 | 35 | 31 | 20
  Hct [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 41 | 38 | 22
  Hct [pre-vacc Normal; post-vacc Below] Month 10 | 6 | 7 | 2
  Hct [pre-vacc Normal ; post-vacc Above] Month 10: number analyzed (Participants) | 41 | 38 | 22
  Hct [pre-vacc Normal ; post-vacc Above] Month 10 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 41 | 38 | 22
  Hct [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 41 | 40 | 22
  Hct [pre-vacc Normal; post-vacc Normal] Month 12 | 32 | 32 | 22
  Hct [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 41 | 40 | 22
  Hct [pre-vacc Normal; post-vacc Below] Month 12 | 9 | 8 | 0
  Hct [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 41 | 40 | 22
  Hct [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 0 | 0
  Hct [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 41 | 40 | 22
  Hct [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 14 | 11 | 2
  Hct [pre-vacc Low; post-vacc Normal] Month 10 | 6 | 4 | 1
  Hct [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 14 | 11 | 2
  Hct [pre-vacc Low; post-vacc Below] Month 10 | 8 | 7 | 1
  Hct [pre-vacc Low ; post-vacc Above] Month 10: number analyzed (Participants) | 14 | 11 | 2
  Hct [pre-vacc Low ; post-vacc Above] Month 10 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 14 | 11 | 2
  Hct [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 13 | 11 | 2
  Hct [pre-vacc Low; post-vacc Normal] Month 12 | 4 | 4 | 1
  Hct [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 13 | 11 | 2
  Hct [pre-vacc Low; post-vacc Below] Month 12 | 9 | 7 | 1
  Hct [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 13 | 11 | 2
  Hct [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  Hct [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 13 | 11 | 2
  Hct [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 10: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 10 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Below] Month 10: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 10 | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 10: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 10 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 10: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 10 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 12: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Normal] Month 12 | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 12: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Below] Month 12 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Above] Month 12: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Above] Month 12 | 0 | 0 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 12: number analyzed (Participants) | 0 | 1 | 0
  Hct [pre-vacc High; post-vacc Missing] Month 12 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 46 | 43 | 21
  Hgb [pre-vacc Normal; post-vacc Normal] Month 10 | 44 | 38 | 21
  Hgb [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 46 | 43 | 21
  Hgb [pre-vacc Normal; post-vacc Below] Month 10 | 2 | 5 | 0
  Hgb [pre-vacc Normal ; post-vacc Above] Month 10: number analyzed (Participants) | 46 | 43 | 21
  Hgb [pre-vacc Normal ; post-vacc Above] Month 10 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 46 | 43 | 21
  Hgb [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 45 | 45 | 21
  Hgb [pre-vacc Normal; post-vacc Normal] Month 12 | 43 | 42 | 21
  Hgb [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 45 | 45 | 21
  Hgb [pre-vacc Normal; post-vacc Below] Month 12 | 2 | 3 | 0
  Hgb [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 45 | 45 | 21
  Hgb [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 0 | 0
  Hgb [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 45 | 45 | 21
  Hgb [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 9 | 7 | 3
  Hgb [pre-vacc Low; post-vacc Normal] Month 10 | 2 | 5 | 1
  Hgb [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 9 | 7 | 3
  Hgb [pre-vacc Low; post-vacc Below] Month 10 | 7 | 2 | 2
  Hgb [pre-vacc Low ; post-vacc Above] Month 10: number analyzed (Participants) | 9 | 7 | 3
  Hgb [pre-vacc Low ; post-vacc Above] Month 10 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 9 | 7 | 3
  Hgb [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 9 | 7 | 3
  Hgb [pre-vacc Low; post-vacc Normal] Month 12 | 4 | 4 | 3
  Hgb [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 9 | 7 | 3
  Hgb [pre-vacc Low; post-vacc Below] Month 12 | 5 | 3 | 0
  Hgb [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 9 | 7 | 3
  Hgb [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  Hgb [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 9 | 7 | 3
  Hgb [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 49 | 49 | 22
  LYM [pre-vacc Normal; post-vacc Normal] Month 10 | 46 | 48 | 21
  LYM [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 49 | 49 | 22
  LYM [pre-vacc Normal; post-vacc Below] Month 10 | 3 | 1 | 0
  LYM [pre-vacc Normal; post-vacc Above] Month 10: number analyzed (Participants) | 49 | 49 | 22
  LYM [pre-vacc Normal; post-vacc Above] Month 10 | 0 | 0 | 1
  LYM [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 49 | 49 | 22
  LYM [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  LYM [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 48 | 51 | 22
  LYM [pre-vacc Normal; post-vacc Normal] Month 12 | 45 | 48 | 21
  LYM [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 48 | 51 | 22
  LYM [pre-vacc Normal; post-vacc Below] Month 12 | 3 | 2 | 1
  LYM [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 48 | 51 | 22
  LYM [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 1 | 0
  LYM [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 48 | 51 | 22
  LYM [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Normal] Month 10 | 4 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 10 | 1 | 0 | 0
  LYM [pre-vacc Low; post-vacc Above] Month 10: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Above] Month 10 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Normal] Month 12 | 3 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Below] Month 12 | 2 | 0 | 0
  LYM [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  LYM [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 5 | 1 | 1
  LYM [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Normal] Month 10: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Normal] Month 10 | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 10: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 10 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Above] Month 10: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Above] Month 10 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Missing] Month 10: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Missing] Month 10 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Normal] Month 12: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Normal] Month 12 | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 12: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Below] Month 12 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Above] Month 12: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Above] Month 12 | 0 | 0 | 0
  LYM [pre-vacc High; post-vacc Missing] Month 12: number analyzed (Participants) | 1 | 0 | 1
  LYM [pre-vacc High; post-vacc Missing] Month 12 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Normal] Month 10: number analyzed (Participants) | 52 | 49 | 24
  MON [pre-vacc Normal; post-vacc Normal] Month 10 | 50 | 48 | 24
  MON [pre-vacc Normal; post-vacc Below] Month 10: number analyzed (Participants) | 52 | 49 | 24
  MON [pre-vacc Normal; post-vacc Below] Month 10 | 2 | 1 | 0
  MON [pre-vacc Normal; post-vacc Above] Month 10: number analyzed (Participants) | 52 | 49 | 24
  MON [pre-vacc Normal; post-vacc Above] Month 10 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Missing] Month 10: number analyzed (Participants) | 52 | 49 | 24
  MON [pre-vacc Normal; post-vacc Missing] Month 10 | 0 | 0 | 0
  MON [pre-vacc Normal; post-vacc Normal] Month 12: number analyzed (Participants) | 51 | 51 | 24
  MON [pre-vacc Normal; post-vacc Normal] Month 12 | 50 | 45 | 24
  MON [pre-vacc Normal; post-vacc Below] Month 12: number analyzed (Participants) | 51 | 51 | 24
  MON [pre-vacc Normal; post-vacc Below] Month 12 | 1 | 5 | 0
  MON [pre-vacc Normal; post-vacc Above] Month 12: number analyzed (Participants) | 51 | 51 | 24
  MON [pre-vacc Normal; post-vacc Above] Month 12 | 0 | 1 | 0
  MON [pre-vacc Normal; post-vacc Missing] Month 12: number analyzed (Participants) | 51 | 51 | 24
  MON [pre-vacc Normal; post-vacc Missing] Month 12 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 10: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 10 | 2 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 10: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 10 | 1 | 0 | 0
  MON [pre-vacc Low; post-vacc Above] Month 10: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Above] Month 10 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 10: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 10 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 12: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Normal] Month 12 | 2 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 12: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Below] Month 12 | 1 | 0 | 0
  MON [pre-vacc Low; post-vacc Above] Month 12: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Above] Month 12 | 0 | 0 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 12: number analyzed (Participants) | 3 | 1 | 0
  MON [pre-vacc Low; post-vacc Missing] Month 12 | 0 | 0 | 0

18. Primary Outcome: Number of Cluster of Differention 4 (CD4+) Cells Per Cubic Millimeter in All HIV+ Subjects at Pre-vaccination (Day 0) and Months 1, 2, 4, 6 and 7
Description: The number of CD4+ cells per cubic millimeter (mm^3) in all HIV+ subjects at pre-vaccination (Day 0) and Months 1, 2, 4, 6 and 7 is reported.
Time Frame: At pre-vaccination (Day 0) and Months 1, 2, 4, 6 and 7
Population: The analysis was performed on the Total Vaccinated cohort, which included all HIV+ vaccinated subjects for whom data were available at the considered time points.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 61 | 59 | 0
cells/mm^3
  Pre-vaccination (Day 0) | 451.0 [310.0 to 596.0] | 458.0 [363.0 to 611.0] |
  Month 1: number analyzed (Participants) | 60 | 57 | 0
  Month 1 | 464.0 [346.0 to 578.5] | 426.0 [352.0 to 584.0] |
  Month 2: number analyzed (Participants) | 58 | 57 | 0
  Month 2 | 436.0 [322.0 to 591.0] | 438.0 [320.0 to 580.0] |
  Month 4: number analyzed (Participants) | 57 | 54 | 0
  Month 4 | 469.0 [346.0 to 596.0] | 423.0 [308.0 to 563.0] |
  Month 6: number analyzed (Participants) | 57 | 54 | 0
  Month 6 | 452.0 [339.0 to 625.0] | 426.0 [334.0 to 550.0] |
  Month 7: number analyzed (Participants) | 56 | 53 | 0
  Month 7 | 419.0 [327.0 to 593.0] | 464.0 [359.0 to 602.0] |

19. Primary Outcome: Number of CD4+ Cells Per Cubic Millimeter in All HIV+ Subjects at Month 10 and Month 12
Description: The number of CD4+ cells per cubic millimeter (mm^3) in all HIV+ subjects at Month 10 and Month 12 is reported.
Time Frame: At Month 10 and Month 12
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 55 | 52 | 0
cells/mm^3
  Month 10: number analyzed (Participants) | 55 | 50 | 0
  Month 10 | 427.0 [347.0 to 621.0] | 442.0 [318.0 to 549.0] |
  Month 12: number analyzed (Participants) | 54 | 52 | 0
  Month 12 | 450.5 [328.0 to 534.0] | 453.0 [332.0 to 636.0] |

20. Primary Outcome: HIV Viral Load in All HIV+ Subjects at Pre-vaccination (Day 0) and Months 1, 2, 4, 6 and 7
Description: The viral load was calculated by estimating the amount of virus in blood samples and it was given in number of Ribonucleic acid copies per milliliter (in log10) [RNA copies/mL (in log10)].
Time Frame: At pre-vaccination (Day 0) and Months 1, 2, 4, 6 and 7
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: RNA copies/mL (in log10)
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 61 | 59 | 0
RNA copies/mL (in log10)
  Pre-vaccination (Day 0) | 4.4 [3.7 to 4.8] | 4.4 [3.7 to 4.7] |
  Month 1: number analyzed (Participants) | 60 | 57 | 0
  Month 1 | 4.4 [3.7 to 4.9] | 4.2 [3.6 to 4.9] |
  Month 2: number analyzed (Participants) | 57 | 57 | 0
  Month 2 | 4.4 [3.6 to 5.1] | 4.6 [4.1 to 4.8] |
  Month 4: number analyzed (Participants) | 57 | 54 | 0
  Month 4 | 4.5 [3.8 to 4.8] | 4.5 [4.0 to 4.9] |
  Month 6: number analyzed (Participants) | 57 | 54 | 0
  Month 6 | 4.6 [3.7 to 5.0] | 4.5 [3.8 to 4.9] |
  Month 7: number analyzed (Participants) | 55 | 53 | 0
  Month 7 | 4.5 [3.8 to 5.0] | 4.5 [3.9 to 4.9] |

21. Primary Outcome: HIV Viral Load in All HIV+ Subjects at Month 10 and Month 12
Description: The viral load was calculated by estimating the amount of virus in blood samples and was given in number of RNA copies/mL (in log 10).
Time Frame: At Month 10 and Month 12
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: RNA copies/mL (in log10)
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 54 | 52 | 0
RNA copies/mL (in log10)
  Month 10: number analyzed (Participants) | 54 | 50 | 0
  Month 10 | 4.5 [4.0 to 4.9] | 4.5 [3.8 to 5.0] |
  Month 12: number analyzed (Participants) | 53 | 52 | 0
  Month 12 | 4.5 [3.8 to 4.9] | 4.5 [3.6 to 4.8] |

22. Primary Outcome: Number of Subjects in Each World Health Organisation (WHO) HIV Clinical Stage by CD4+ Cell Count Category at Baseline in All HIV+ Subjects at Months 1, 2, 4, 6 and 7
Description: CD4+ cell count categories, at baseline, assessed were (i) below (<) 200 CD4+ cells per cubic millimeter (mm^3), (ii) between 200 and 500 CD4+ cells/mm^3 and (iii) above 500 CD4+ cells/mm^3. WHO classification of HIV-associated clinical disease: 1 = Asymptomatic HIV-associated symptoms = WHO clinical stage 1; 2 = Mild HIV-associated symptoms = WHO clinical stage 2; 3 = Advanced HIV-associated symptoms = WHO clinical stage 3; 4 = Severe HIV-associated symptoms = WHO clinical stage 4.
Time Frame: At Months 1, 2, 4, 6 and 7
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 60 | 57 | 0
Participants
  <200 CD4+cells/mm^3 [stage 1] Month 1: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 1] Month 1 | 2 | 1 |
  <200 CD4+cells/mm^3 [stage 2] Month 1: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 2] Month 1 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 3] Month 1: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 3] Month 1 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 4] Month 1: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 4] Month 1 | 0 | 0 |
  200-500 CD4+cells/mm^3 [stage 1] Month 1: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 1] Month 1 | 31 | 33 |
  200-500 CD4+cells/mm^3 [stage 2] Month 1: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 2] Month 1 | 2 | 2 |
  200-500 CD4+cells/mm^3 [stage 3] Month 1: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 3] Month 1 | 2 | 1 |
  200-500 CD4+cells/mm^3 [stage 4] Month 1: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 4] Month 1 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 1] Month 1: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 1] Month 1 | 23 | 20 |
  >500 CD4+cells/mm^3 [stage 2] Month 1: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 2] Month 1 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 3] Month 1: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 3] Month 1 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 4] Month 1: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 4] Month 1 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 1] Month 2: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 1] Month 2 | 2 | 1 |
  <200 CD4+cells/mm^3 [stage 2] Month 2: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 2] Month 2 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 3] Month 2: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 3] Month 2 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 4] Month 2: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 4] Month 2 | 0 | 0 |
  200-500 CD4+cells/mm^3 [stage 1] Month 2: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 1] Month 2 | 30 | 33 |
  200-500 CD4+cells/mm^3 [stage 2] Month 2: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 2] Month 2 | 2 | 3 |
  200-500 CD4+cells/mm^3 [stage 3] Month 2: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 3] Month 2 | 2 | 1 |
  200-500 CD4+cells/mm^3 [stage 4] Month 2: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 4] Month 2 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 1] Month 2: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 1] Month 2 | 22 | 19 |
  >500 CD4+cells/mm^3 [stage 2] Month 2: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 2] Month 2 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 3] Month 2: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 3] Month 2 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 4] Mth 2: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 4] Mth 2 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 1] Month 4: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 1] Month 4 | 2 | 1 |
  <200 CD4+cells/mm^3 [stage 2] Month 4: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 2] Month 4 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 3] Month 4: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 3] Month 4 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 4] Month 4: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 4] Month 4 | 0 | 0 |
  200-500 CD4+cells/mm^3 [stage 1] Month 4: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 1] Month 4 | 28 | 27 |
  200-500 CD4+cells/mm^3 [stage 2] Month 4: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 2] Month 4 | 2 | 1 |
  200-500 CD4+cells/mm^3 [stage 3] Month 4: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 3] Month 4 | 2 | 5 |
  200-500 CD4+cells/mm^3 [stage 4] Month 4: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 4] Month 4 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 1] Month 4: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 1] Month 4 | 23 | 20 |
  >500 CD4+cells/mm^3 [stage 2] Month 4: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 2] Month 4 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 3] Month 4: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 3] Month 4 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 4] Month 4: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 4] Month 4 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 1] Month 6: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 1] Month 6 | 2 | 1 |
  <200 CD4+cells/mm^3 [stage 2] Month 6: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 2] Month 6 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 3] Month 6: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 3] Month 6 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 4] Month 6: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 4] Month 6 | 0 | 0 |
  200-500 CD4+cells/mm^3 [stage 1] Month 6: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 1] Month 6 | 28 | 28 |
  200-500 CD4+cells/mm^3 [stage 2] Month 6: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 2] Month 6 | 2 | 1 |
  200-500 CD4+cells/mm^3 [stage 3] Month 6: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 3] Month 6 | 2 | 5 |
  200-500 CD4+cells/mm^3 [stage 4] Month 6: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 4] Month 6 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 1] Month 6: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 1] Month 6 | 23 | 19 |
  >500 CD4+cells/mm^3 [stage 2] Month 6: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 2] Month 6 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 3] Month 6: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 3] Month 6 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 4] Month 6: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 4] Month 6 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 1] Month 7: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 1] Month 7 | 2 | 1 |
  <200 CD4+cells/mm^3 [stage 2] Month 7: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 2] Month 7 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 3] Month 7: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 3] Month 7 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 4] Month 7: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 4] Month 7 | 0 | 0 |
  200-500 CD4+cells/mm^3 [stage 1] Month 7: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 1] Month 7 | 28 | 28 |
  200-500 CD4+cells/mm^3 [stage 2] Month 7: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 2] Month 7 | 2 | 0 |
  200-500 CD4+cells/mm^3 [stage 3] Month 7: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 3] Month 7 | 2 | 4 |
  200-500 CD4+cells/mm^3 [stage 4] Month 7: number analyzed (Participants) | 35 | 36 | 0
  200-500 CD4+cells/mm^3 [stage 4] Month 7 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 1] Month 7: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 1] Month 7 | 21 | 19 |
  >500 CD4+cells/mm^3 [stage 2] Month 7: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 2] Month 7 | 1 | 1 |
  >500 CD4+cells/mm^3 [stage 3] Month 7: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 3] Month 7 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 4] Month 7: number analyzed (Participants) | 23 | 20 | 0
  >500 CD4+cells/mm^3 [stage 4] Month 7 | 0 | 0 |

23. Primary Outcome: Number of Subjects in Each World Health Organisation (WHO) HIV Clinical Stage by CD4+ Cell Count Category at Baseline in All HIV+ Subjects at Month 10 and Month 12
Description: CD4+ cell count categories, at baseline, assessed were: (i) below (<) 200 CD4+ cells per cubic millimeter (mm^3), (ii) between 200 and 500 CD4+ cells/mm^3 and (iii) above (>) 500 CD4+ cells/mm^3. WHO classification of HIV-associated clinical disease: 1 = Asymptomatic HIV-associated symptoms = WHO clinical stage 1; 2 = Mild HIV-associated symptoms = WHO clinical stage 2; 3 = Advanced HIV-associated symptoms = WHO clinical stage 3; 4 = Severe HIV-associated symptoms = WHO clinical stage 4.
Time Frame: At Month 10 and Month 12
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 55 | 52 | 0
Participants
  <200 CD4+cells/mm^3 [stage 1] Month 10: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 1] Month 10 | 1 | 1 |
  <200 CD4+cells/mm^3 [stage 2] Month 10: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 2] Month 10 | 1 | 0 |
  <200 CD4+cells/mm^3 [stage 3] Month 10: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 3] Month 10 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 4] Month 10: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 4] Month 10 | 0 | 0 |
  200-500 CD4+cells/mm^3 [stage 1] Month 10: number analyzed (Participants) | 31 | 30 | 0
  200-500 CD4+cells/mm^3 [stage 1] Month 10 | 26 | 25 |
  200-500 CD4+cells/mm^3 [stage 2] Month 10: number analyzed (Participants) | 31 | 30 | 0
  200-500 CD4+cells/mm^3 [stage 2] Month 10 | 1 | 0 |
  200-500 CD4+cells/mm^3 [stage 3] Month 10: number analyzed (Participants) | 31 | 30 | 0
  200-500 CD4+cells/mm^3 [stage 3] Month 10 | 4 | 4 |
  200-500 CD4+cells/mm^3 [stage 4] Month 10: number analyzed (Participants) | 31 | 30 | 0
  200-500 CD4+cells/mm^3 [stage 4] Month 10 | 0 | 1 |
  >500 CD4+cells/mm^3 [stage 1] Month 10: number analyzed (Participants) | 22 | 19 | 0
  >500 CD4+cells/mm^3 [stage 1] Month 10 | 21 | 18 |
  >500 CD4+cells/mm^3 [stage 2] Month 10: number analyzed (Participants) | 22 | 19 | 0
  >500 CD4+cells/mm^3 [stage 2] Month 10 | 1 | 1 |
  >500 CD4+cells/mm^3 [stage 3] Month 10: number analyzed (Participants) | 22 | 19 | 0
  >500 CD4+cells/mm^3 [stage 3] Month 10 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 4] Month 10: number analyzed (Participants) | 22 | 19 | 0
  >500 CD4+cells/mm^3 [stage 4] Month 10 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 1] Month 12: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 1] Month 12 | 0 | 1 |
  <200 CD4+cells/mm^3 [stage 2] Month 12: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 2] Month 12 | 2 | 0 |
  <200 CD4+cells/mm^3 [stage 3] Month 12: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 3] Month 12 | 0 | 0 |
  <200 CD4+cells/mm^3 [stage 4] Month 12: number analyzed (Participants) | 2 | 1 | 0
  <200 CD4+cells/mm^3 [stage 4] Month 12 | 0 | 0 |
  200-500 CD4+cells/mm^3 [stage 1] Month 12: number analyzed (Participants) | 31 | 32 | 0
  200-500 CD4+cells/mm^3 [stage 1] Month 12 | 24 | 23 |
  200-500 CD4+cells/mm^3 [stage 2] Month 12: number analyzed (Participants) | 31 | 32 | 0
  200-500 CD4+cells/mm^3 [stage 2] Month 12 | 3 | 2 |
  200-500 CD4+cells/mm^3 [stage 3] Month 12: number analyzed (Participants) | 31 | 32 | 0
  200-500 CD4+cells/mm^3 [stage 3] Month 12 | 4 | 6 |
  200-500 CD4+cells/mm^3 [stage 4] Month 12: number analyzed (Participants) | 31 | 32 | 0
  200-500 CD4+cells/mm^3 [stage 4] Month 12 | 0 | 1 |
  >500 CD4+cells/mm^3 [stage 1] Month 12: number analyzed (Participants) | 21 | 19 | 0
  >500 CD4+cells/mm^3 [stage 1] Month 12 | 20 | 17 |
  >500 CD4+cells/mm^3 [stage 2] Month 12: number analyzed (Participants) | 21 | 19 | 0
  >500 CD4+cells/mm^3 [stage 2] Month 12 | 1 | 2 |
  >500 CD4+cells/mm^3 [stage 3] Month 12: number analyzed (Participants) | 21 | 19 | 0
  >500 CD4+cells/mm^3 [stage 3] Month 12 | 0 | 0 |
  >500 CD4+cells/mm^3 [stage 4] Month 12: number analyzed (Participants) | 21 | 19 | 0
  >500 CD4+cells/mm^3 [stage 4] Month 12 | 0 | 0 |

24. Primary Outcome: Number of Seroconverted Subjects for HPV-16 and HPV-18 Antibodies at Pre-vaccination (Day 0) and Months 2 and 7
Description: Seroconversion is defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies (anti-HPV-16 titers ≥ 8 EL.U/mL and anti-HPV-18 titers ≥ 7 EL.U/mL) in the serum of subjects seronegative before vaccination. A seronegative subject is a subject whose antibody titers are below the cut-off value. Due to the high proportion of initially seropositive subjects in the study population, seroconversion rates were considered for all subjects in the According-to-Protocol (ATP) cohort for immunogenicity regardless of baseline serostatus.
Time Frame: At pre-vaccination (Day 0) and Months 2 and 7
Population: The analysis was performed on the ATP cohort for immunogenicity (Month 7), which included all evaluable subjects up to Month 7 for whom immunogenicity data were available at the considered time points. This included subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component post-vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 43 | 40 | 24
Participants
  anti-HPV-16, At Day 0: number analyzed (Participants) | 42 | 40 | 24
  anti-HPV-16, At Day 0 | 35 | 30 | 14
  anti-HPV-16, At Month 2: number analyzed (Participants) | 41 | 40 | 24
  anti-HPV-16, At Month 2 | 41 | 31 | 24
  anti-HPV-16, At Month 7: number analyzed (Participants) | 42 | 40 | 24
  anti-HPV-16, At Month 7 | 42 | 31 | 24
  anti-HPV-18, At Day 0 | 27 | 24 | 11
  anti-HPV-18, At Month 2: number analyzed (Participants) | 42 | 40 | 24
  anti-HPV-18, At Month 2 | 42 | 26 | 24
  anti-HPV-18, At Month 7 | 43 | 25 | 24

25. Primary Outcome: Number of Seroconverted Subjects for HPV-16 and HPV-18 Antibodies at Month 12
Description: Seroconversion is defined as the appearance of anti-HPV-16 and/or anti-HPV-18 antibodies (anti-HPV-16 titers ≥ 8 ELISA units per milliliter (EL.U/mL) and anti-HPV-18 titers ≥ 7 EL.U/mL) in the serum of subjects seronegative before vaccination. A seronegative subject is a subject whose antibody titers are below the cut-off value. Due to the high proportion of initially seropositive subjects in the study population, seroconversion rates were considered for all subjects in the ATP cohort for immunogenicity regardless of baseline serostatus.
Time Frame: At Month 12
Population: The analysis was performed on ATP cohort for immunogenicity (Month 12), which included all evaluable subjects up to Month 12 for whom immunogenicity data were available at the considered time points. This included subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component post-vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 42 | 37 | 22
Participants
  anti-HPV-16, At Month 12: number analyzed (Participants) | 41 | 37 | 22
  anti-HPV-16, At Month 12 | 41 | 28 | 22
  anti-HPV-18, At Month 12 | 42 | 24 | 22

26. Primary Outcome: Concentrations for HPV-16 and HPV-18 Antibodies at Pre-vaccination (Day 0) and Months 2 and 7
Description: Concentrations are expressed as geometric mean antibody concentrations (GMCs) and are given in EL.U/mL. The antibody concentrations against HPV-16 and HPV-18 were determined by Enzyme-linked immunosorbent assay (ELISA). The cut-off values of the assay are 8 EL.U/mL for anti-HPV-16 and 7 EL.U/mL for anti-HPV-18.
Time Frame: At pre-vaccination (Day 0) and Months 2 and 7
Population: as for outcome 24
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 43 | 40 | 24
EL.U/mL
  anti-HPV-16, At Day 0: number analyzed (Participants) | 42 | 40 | 24
  anti-HPV-16, At Day 0 | 29.7 [20.1 to 43.7] | 25.7 [16.6 to 39.9] | 21.8 [10.9 to 43.3]
  anti-HPV-16, At Month 2: number analyzed (Participants) | 41 | 40 | 24
  anti-HPV-16, At Month 2 | 2245.2 [1634.2 to 3084.5] | 32.9 [19.3 to 56.0] | 6166.8 [4079.5 to 9322.2]
  anti-HPV-16, At Month 7: number analyzed (Participants) | 42 | 40 | 24
  anti-HPV-16, At Month 7 | 3583.1 [2759.9 to 4651.9] | 27.2 [17.6 to 42.0] | 7871.9 [6185.3 to 10018.4]
  anti-HPV-18, At Day 0 | 13.2 [9.0 to 19.3] | 12.5 [8.2 to 19.1] | 11.1 [5.8 to 21.2]
  anti-HPV-18, At Month 2: number analyzed (Participants) | 42 | 40 | 24
  anti-HPV-18, At Month 2 | 1339.3 [901.6 to 1989.5] | 16.9 [10.1 to 28.3] | 2380.2 [1718.7 to 3296.2]
  anti-HPV-18, At Month 7 | 1952.1 [1466.3 to 2598.7] | 14.5 [9.2 to 22.9] | 3755.3 [2608.4 to 5406.5]

27. Primary Outcome: Concentrations for HPV-16 and HPV-18 Antibodies at Month 12
Description: as for outcome 26
Time Frame: At Month 12
Population: The analysis was performed on the ATP cohort for immunogenicity (Month 12), which included all evaluable subjects up to Month 12 for whom immunogenicity data were available at the considered time points. This included subjects for whom assay results were available for antibodies against at least 1 study vaccine antigen component post-vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 42 | 37 | 22
EL.U/mL
  anti-HPV-16, At Month 12: number analyzed (Participants) | 41 | 37 | 22
  anti-HPV-16, At Month 12 | 748.1 [520.0 to 1076.3] | 20.7 [13.9 to 30.9] | 2793.6 [2087.8 to 3738.0]
  anti-HPV-18, At Month 12 | 343.1 [236.2 to 498.2] | 13.0 [8.5 to 19.7] | 1021.3 [627.4 to 1662.6]

28. Primary Outcome: Cell Mediated Immune (CMI) Response (B-cell Responses) Related to HPV 16/18 Virus-like Particles (VLPs) Measured by Flow Cytometry at Day 0
Description: The CMI response is expressed by the number of subjects with B-cell response to VLP-16 and VLP-18 above (>) 0 as measured by Flow cytometry.
Time Frame: At pre-vaccination (Day 0)
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 42 | 37 | 22
Participants
  VLP-16, =0 | 8 | 13 | 10
  VLP-16, >0 | 14 | 13 | 6
  VLP-16, Missing | 20 | 11 | 6
  VLP-18, =0 | 5 | 15 | 6
  VLP-18, >0 | 16 | 11 | 10
  VLP-18, Missing | 21 | 11 | 6

29. Primary Outcome: CMI B-cell Responses Related to HPV 16/18 Virus-like Particles (VLPs) Measured by Flow Cytometry at Month 2
Description: as for outcome 28
Time Frame: At Month 2
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 42 | 37 | 22
Participants
  VLP-16, =0 | 8 | 9 | 2
  VLP-16, >0 | 20 | 7 | 11
  VLP-16, Missing | 14 | 21 | 9
  VLP-18, =0 | 11 | 9 | 2
  VLP-18, >0 | 17 | 8 | 11
  VLP-18, Missing | 14 | 20 | 9

30. Primary Outcome: CMI B-cell Responses Related to HPV 16/18 Virus-like Particles (VLPs) Measured by Flow Cytometry at Month 7
Description: as for outcome 28
Time Frame: At Month 7
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 42 | 37 | 22
Participants
  VLP-16, =0 | 2 | 9 | 1
  VLP-16, >0 | 24 | 16 | 21
  VLP-16, Missing | 16 | 12 | 0
  VLP-18, =0 | 0 | 15 | 1
  VLP-18, >0 | 25 | 11 | 19
  VLP-18, Missing | 17 | 11 | 2

31. Primary Outcome: CMI B-cell Responses Related to HPV 16/18 Virus-like Particles (VLPs) Measured by Flow Cytometry at Month 12
Description: as for outcome 28
Time Frame: At Month 12
Population: as for outcome 27
Measure: Count of Participants; unit: Participants
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 42 | 37 | 22
Participants
  VLP-16, =0 | 8 | 9 | 2
  VLP-16, >0 | 21 | 16 | 18
  VLP-16, Missing | 13 | 12 | 2
  VLP-18, =0 | 13 | 10 | 3
  VLP-18, >0 | 13 | 14 | 15
  VLP-18, Missing | 16 | 13 | 4

32. Primary Outcome: CMI Response (T-cell Responses) Related to HPV-16 and HPV-18 Measured by Intracellular Cytokine Staining (ICS)
Description: The CMI response is the measure of the cytokines production [i.e. Cluster of Differentiation 40 Ligand (CD40L), Interferon gamma (IFN-γ), interleukin-2 (IL-2) and tumor necrosis factor alpha (TNF-α)] by HPV-antigen specific T lymphocytes and measured by Intracellular Cytokine Staining (ICS) assay. The results were expressed as a frequency of positive CD4 or CD8 T-cell producing at least 1 cytokine within the CD4 or CD8 T-cell sub-population. All doubles = T cell expressing at least 2 cytokines.
Time Frame: At pre-vaccination (Day 0) and at Months 2, 7 and 12
Population: as for outcome 27
Measure: Geometric Mean (Inter-Quartile Range); unit: T cells/million cells
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
Number analyzed (Participants) | 36 | 32 | 18
T cells/million cells
  CD4-ALL DOUBLES [HPV-16], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-ALL DOUBLES [HPV-16], At Day 0 | 256.0 [119.0 to 390.0] | 154.0 [96.0 to 235.0] | 259.0 [160.0 to 377.0]
  CD4-ALL DOUBLES [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-ALL DOUBLES [HPV-16], At Month 2 | 4082.0 [2997.0 to 6209.0] | 154.5 [94.0 to 293.0] | 1691.0 [1247.0 to 2809.0]
  CD4-ALL DOUBLES [HPV-16], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4-ALL DOUBLES [HPV-16], At Month 7 | 4717.5 [2050.5 to 9242.5] | 177.5 [106.0 to 302.0] | 3121.5 [1726.0 to 4538.0]
  CD4-ALL DOUBLES [HPV-16], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4-ALL DOUBLES [HPV-16], At Month 12 | 3063.5 [1294.0 to 5294.5] | 184.5 [136.0 to 326.5] | 2490.0 [1247.0 to 4499.0]
  CD4-ALL DOUBLES [HPV-18], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-ALL DOUBLES [HPV-18], At Day 0 | 218.0 [131.0 to 281.0] | 114.0 [82.0 to 188.0] | 273.0 [135.0 to 387.0]
  CD4-ALL DOUBLES [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-ALL DOUBLES [HPV-18], At Month 2 | 2658.0 [1157.0 to 4197.0] | 156.5 [98.0 to 231.0] | 1065.0 [624.0 to 1681.0]
  CD4-ALL DOUBLES [HPV-18], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4-ALL DOUBLES [HPV-18], At Month 7 | 2917.5 [1365.0 to 5976.0] | 143.5 [88.5 to 227.5] | 1834.0 [973.0 to 2827.0]
  CD4-ALL DOUBLES [HPV-18], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4-ALL DOUBLES [HPV-18], At Month 12 | 1694.5 [783.0 to 3401.0] | 220.0 [121.0 to 285.5] | 1783.0 [939.0 to 2891.0]
  CD4-CD40L [HPV-16], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-CD40L [HPV-16], At Day 0 | 200.0 [97.0 to 277.0] | 101.0 [50.0 to 170.0] | 208.0 [119.0 to 239.0]
  CD4-CD40L [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-CD40L [HPV-16], At Month 2 | 3940.0 [2653.0 to 5999.0] | 125.5 [82.0 to 229.0] | 1437.0 [1165.0 to 2649.0]
  CD4-CD40L [HPV-16], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4-CD40L [HPV-16], At Month 7 | 3400.5 [1743.0 to 6893.0] | 143.5 [50.0 to 182.0] | 2303.0 [1483.0 to 3871.0]
  CD4-CD40L [HPV-16], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4-CD40L [HPV-16], At Month 12 | 2569.0 [1209.5 to 4946.5] | 162.5 [81.5 to 320.0] | 2201.0 [930.0 to 4090.0]
  CD4-CD40L [HPV-18], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-CD40L [HPV-18], At Day 0 | 150.0 [110.0 to 225.0] | 98.0 [45.0 to 147.0] | 222.0 [82.0 to 306.0]
  CD4-CD40L [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-CD40L [HPV-18], At Month 2 | 2467.0 [911.0 to 3549.0] | 142.5 [75.0 to 195.0] | 974.0 [509.0 to 1598.0]
  CD4-CD40L [HPV-18], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4-CD40L [HPV-18], At Month 7 | 2247.5 [1154.0 to 4510.0] | 108.5 [50.5 to 185.0] | 1524.5 [706.0 to 2327.0]
  CD4-CD40L [HPV-18], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4-CD40L [HPV-18], At Month 12 | 1484.0 [739.5 to 3045.0] | 178.0 [90.0 to 250.0] | 1587.0 [782.0 to 2596.0]
  CD4-IFN-γ [HPV-16], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-IFN-γ [HPV-16], At Day 0 | 57.0 [31.0 to 161.0] | 57.0 [7.0 to 85.0] | 66.0 [50.0 to 102.0]
  CD4-IFN-γ [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-IFN-γ [HPV-16], At Month 2 | 1748.0 [890.0 to 2632.0] | 50.0 [7.0 to 85.0] | 760.0 [535.0 to 956.0]
  CD4- IFN-γ [HPV-16], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4- IFN-γ [HPV-16], At Month 7 | 1807.0 [741.5 to 3483.0] | 51.0 [7.0 to 111.0] | 900.5 [763.0 to 1718.0]
  CD4- IFN-γ [HPV-16], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4- IFN-γ [HPV-16], At Month 12 | 735.0 [365.0 to 1290.5] | 49.5 [19.0 to 97.5] | 592.0 [320.0 to 895.0]
  CD4-IFN-γ [HPV-18], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-IFN-γ [HPV-18], At Day 0 | 25.0 [7.0 to 99.0] | 40.0 [7.0 to 58.0] | 54.0 [34.0 to 72.0]
  CD4-IFN-γ [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-IFN-γ [HPV-18], At Month 2 | 1045.0 [422.0 to 1619.0] | 43.5 [7.0 to 77.0] | 407.0 [285.0 to 532.0]
  CD4- IFN-γ [HPV-18], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4- IFN-γ [HPV-18], At Month 7 | 915.0 [453.0 to 2156.5] | 31.5 [7.0 to 68.5] | 626.5 [415.0 to 917.0]
  CD4- IFN-γ [HPV-18], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4- IFN-γ [HPV-18], At Month 12 | 341.5 [226.5 to 1052.0] | 39.0 [7.0 to 91.5] | 436.0 [291.0 to 587.0]
  CD4-IL-2 [HPV-16], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-IL-2 [HPV-16], At Day 0 | 187.0 [97.0 to 285.0] | 104.0 [42.0 to 150.0] | 176.0 [105.0 to 313.0]
  CD4-IL-2 [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-IL-2 [HPV-16], At Month 2 | 3716.0 [2951.0 to 5879.0] | 79.0 [44.0 to 148.0] | 1601.0 [1030.0 to 2493.0]
  CD4- IL-2 [HPV-16], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4- IL-2 [HPV-16], At Month 7 | 4329.0 [1939.0 to 8847.0] | 113.5 [52.5 to 175.0] | 2830.5 [1509.0 to 4251.0]
  CD4- IL-2 [HPV-16], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4- IL-2 [HPV-16], At Month 12 | 2946.0 [983.5 to 4840.5] | 135.5 [62.0 to 235.5] | 2366.0 [1075.0 to 4397.0]
  CD4-IL-2 [HPV-18], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-IL-2 [HPV-18], At Day 0 | 132.0 [50.0 to 225.0] | 76.0 [43.0 to 106.0] | 206.0 [109.0 to 301.0]
  CD4-IL-2 [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-IL-2 [HPV-18], At Month 2 | 2527.0 [1153.0 to 3850.0] | 103.5 [55.0 to 158.0] | 921.0 [587.0 to 1428.0]
  CD4- IL-2 [HPV-18], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4- IL-2 [HPV-18], At Month 7 | 2664.0 [1258.0 to 5289.0] | 87.5 [57.0 to 153.5] | 1572.5 [900.0 to 2678.0]
  CD4- IL-2 [HPV-18], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4- IL-2 [HPV-18], At Month 12 | 1533.5 [713.5 to 3229.0] | 134.0 [57.0 to 206.5] | 1633.0 [741.0 to 2787.0]
  CD4-TNF-α [HPV-16], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-TNF-α [HPV-16], At Day 0 | 148.0 [61.0 to 226.0] | 132.0 [50.0 to 221.0] | 185.0 [127.0 to 261.0]
  CD4-TNF-α [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-TNF-α [HPV-16], At Month 2 | 3131.0 [1811.0 to 4864.0] | 105.0 [55.0 to 215.0] | 1332.0 [980.0 to 1894.0]
  CD4-TNF-α [HPV-16], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4-TNF-α [HPV-16], At Month 7 | 4315.0 [1815.5 to 8347.5] | 154.0 [58.0 to 247.5] | 2479.0 [1426.0 to 3988.0]
  CD4-TNF-α [HPV-16], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4-TNF-α [HPV-16], At Month 12 | 2662.5 [1088.0 to 4675.0] | 135.5 [81.5 to 257.0] | 2133.0 [1125.0 to 4064.0]
  CD4-TNF-α [HPV-18], At Day 0: number analyzed (Participants) | 33 | 29 | 15
  CD4-TNF-α [HPV-18], At Day 0 | 150.0 [92.0 to 211.0] | 84.0 [72.0 to 148.0] | 229.0 [65.0 to 295.0]
  CD4-TNF-α [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD4-TNF-α [HPV-18], At Month 2 | 2319.0 [1065.0 to 3666.0] | 94.5 [56.0 to 173.0] | 982.0 [505.0 to 1198.0]
  CD4-TNF-α [HPV-18], At Month 7: number analyzed (Participants) | 32 | 32 | 18
  CD4-TNF-α [HPV-18], At Month 7 | 2689.0 [1236.5 to 5303.5] | 109.0 [58.5 to 168.5] | 1526.5 [869.0 to 2682.0]
  CD4-TNF-α [HPV-18], At Month 12: number analyzed (Participants) | 36 | 28 | 13
  CD4-TNF-α [HPV-18], At Month 12 | 1542.5 [627.5 to 3175.5] | 138.0 [59.5 to 198.5] | 1650.0 [860.0 to 2541.0]
  CD8-ALL DOUBLES [HPV-16], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-ALL DOUBLES [HPV-16], At Day 0 | 43.0 [16.0 to 79.0] | 40.0 [11.0 to 58.0] | 26.0 [11.0 to 73.0]
  CD8-ALL DOUBLES [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8-ALL DOUBLES [HPV-16], At Month 2 | 65.0 [34.0 to 107.0] | 40.5 [11.0 to 90.0] | 48.0 [34.0 to 118.0]
  CD8-ALL DOUBLES [HPV-16], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-ALL DOUBLES [HPV-16], At Month 7 | 38.0 [24.5 to 94.0] | 32.5 [11.0 to 76.0] | 48.0 [26.0 to 71.0]
  CD8-ALL DOUBLES [HPV-16], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-ALL DOUBLES [HPV-16], At Month 12 | 53.5 [11.0 to 118.5] | 37.0 [11.0 to 72.0] | 45.0 [11.0 to 58.0]
  CD8-ALL DOUBLES [HPV-18], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-ALL DOUBLES [HPV-18], At Day 0 | 51.0 [29.5 to 89.0] | 11.0 [11.0 to 58.0] | 31.0 [11.0 to 63.0]
  CD8-ALL DOUBLES [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8-ALL DOUBLES [HPV-18], At Month 2 | 65.0 [11.0 to 85.0] | 39.5 [11.0 to 91.0] | 62.0 [32.0 to 85.0]
  CD8-ALL DOUBLES [HPV-18], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-ALL DOUBLES [HPV-18], At Month 7 | 40.0 [15.5 to 100.0] | 35.5 [11.0 to 63.0] | 44.0 [11.0 to 74.0]
  CD8-ALL DOUBLES [HPV-18], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-ALL DOUBLES [HPV-18], At Month 12 | 39.5 [11.0 to 128.5] | 35.0 [11.0 to 75.0] | 21.0 [11.0 to 47.0]
  CD8-CD40L [HPV-16], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-CD40L [HPV-16], At Day 0 | 7.0 [7.0 to 31.0] | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 34.0]
  CD8-CD40L [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8-CD40L [HPV-16], At Month 2 | 28.0 [7.0 to 55.0] | 7.0 [7.0 to 27.0] | 7.0 [7.0 to 44.0]
  CD8-CD40L [HPV-16], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-CD40L [HPV-16], At Month 7 | 26.5 [7.0 to 38.5] | 7.0 [7.0 to 20.0] | 24.0 [7.0 to 49.0]
  CD8-CD40L [HPV-16], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-CD40L [HPV-16], At Month 12 | 7.0 [7.0 to 15.5] | 7.0 [7.0 to 32.0] | 7.0 [7.0 to 7.0]
  CD8-CD40L [HPV-18], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-CD40L [HPV-18], At Day 0 | 18.5 [7.0 to 36.5] | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 27.0]
  CD8- CD40L [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8- CD40L [HPV-18], At Month 2 | 7.0 [7.0 to 42.0] | 7.0 [7.0 to 43.0] | 38.0 [7.0 to 60.0]
  CD8-CD40L [HPV-18], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-CD40L [HPV-18], At Month 7 | 7.0 [7.0 to 29.0] | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 57.0]
  CD8-CD40L [HPV-18], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-CD40L [HPV-18], At Month 12 | 7.0 [7.0 to 23.0] | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0]
  CD8-IFN-γ [HPV-16], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-IFN-γ [HPV-16], At Day 0 | 35.5 [7.0 to 73.5] | 25.0 [7.0 to 54.0] | 7.0 [7.0 to 42.0]
  CD8-IFN-γ [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8-IFN-γ [HPV-16], At Month 2 | 39.0 [24.0 to 103.0] | 7.0 [7.0 to 80.0] | 39.0 [22.0 to 62.0]
  CD8-IFN-γ [HPV-16], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-IFN-γ [HPV-16], At Month 7 | 25.0 [7.0 to 76.0] | 23.5 [7.0 to 66.0] | 28.5 [7.0 to 55.0]
  CD8-IFN-γ [HPV-16], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-IFN-γ [HPV-16], At Month 12 | 47.5 [7.0 to 106.0] | 28.5 [7.0 to 43.0] | 26.0 [7.0 to 50.0]
  CD8-IFN-γ [HPV-18], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-IFN-γ [HPV-18], At Day 0 | 39.0 [7.0 to 85.0] | 7.0 [7.0 to 47.0] | 9.0 [7.0 to 41.0]
  CD8-IFN-γ [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8-IFN-γ [HPV-18], At Month 2 | 37.0 [7.0 to 78.0] | 27.5 [7.0 to 84.0] | 53.0 [23.0 to 68.0]
  CD8-IFN-γ [HPV-18], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-IFN-γ [HPV-18], At Month 7 | 33.0 [8.5 to 82.0] | 22.0 [7.0 to 59.0] | 38.0 [7.0 to 59.0]
  CD8-IFN-γ [HPV-18], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-IFN-γ [HPV-18], At Month 12 | 29.0 [7.0 to 96.5] | 31.0 [7.0 to 54.0] | 7.0 [7.0 to 23.0]
  CD8-IL-2 [HPV-16], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-IL-2 [HPV-16], At Day 0 | 7.0 [7.0 to 29.0] | 7.0 [7.0 to 25.0] | 7.0 [7.0 to 34.0]
  CD8-IL-2 [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8-IL-2 [HPV-16], At Month 2 | 24.0 [7.0 to 35.0] | 20.0 [7.0 to 34.0] | 32.0 [7.0 to 62.0]
  CD8-IL-2 [HPV-16], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-IL-2 [HPV-16], At Month 7 | 20.5 [7.0 to 33.0] | 7.0 [7.0 to 7.0] | 28.5 [7.0 to 55.0]
  CD8-IL-2 [HPV-16], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-IL-2 [HPV-16], At Month 12 | 7.0 [7.0 to 38.5] | 7.5 [7.0 to 33.0] | 7.0 [7.0 to 27.0]
  CD8-IL-2 [HPV-18], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-IL-2 [HPV-18], At Day 0 | 7.0 [7.0 to 30.5] | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 32.0]
  CD8-IL-2 [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8-IL-2 [HPV-18], At Month 2 | 7.0 [7.0 to 37.0] | 7.0 [7.0 to 24.0] | 11.0 [7.0 to 44.0]
  CD8-IL-2 [HPV-18], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-IL-2 [HPV-18], At Month 7 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 7.0] | 17.5 [7.0 to 41.0]
  CD8-IL-2 [HPV-18], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-IL-2 [HPV-18], At Month 12 | 7.0 [7.0 to 7.0] | 7.0 [7.0 to 17.0] | 7.0 [7.0 to 38.0]
  CD8-TNF-α [HPV-16], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-TNF-α [HPV-16], At Day 0 | 26.0 [7.0 to 71.0] | 34.0 [7.0 to 54.0] | 7.0 [7.0 to 36.0]
  CD8-TNF-α [HPV-16], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8-TNF-α [HPV-16], At Month 2 | 34.0 [7.0 to 52.0] | 28.5 [7.0 to 65.0] | 30.0 [7.0 to 55.0]
  CD8-TNF-α [HPV-16], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-TNF-α [HPV-16], At Month 7 | 25.5 [7.0 to 53.5] | 15.5 [7.0 to 66.0] | 28.5 [7.0 to 50.0]
  CD8-TNF-α [HPV-16], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-TNF-α [HPV-16], At Month 12 | 35.5 [7.0 to 97.0] | 9.0 [7.0 to 38.0] | 26.0 [7.0 to 50.0]
  CD8-TNF-α [HPV-18], At Day 0: number analyzed (Participants) | 32 | 29 | 15
  CD8-TNF-α [HPV-18], At Day 0 | 21.5 [7.0 to 55.0] | 7.0 [7.0 to 46.0] | 7.0 [7.0 to 41.0]
  CD8-TNF-α [HPV-18], At Month 2: number analyzed (Participants) | 29 | 26 | 17
  CD8-TNF-α [HPV-18], At Month 2 | 38.0 [7.0 to 66.0] | 7.0 [7.0 to 54.0] | 28.0 [7.0 to 50.0]
  CD8-TNF-α [HPV-18], At Month 7: number analyzed (Participants) | 32 | 30 | 18
  CD8-TNF-α [HPV-18], At Month 7 | 28.5 [7.0 to 73.5] | 25.5 [7.0 to 57.0] | 22.0 [7.0 to 59.0]
  CD8-TNF-α [HPV-18], At Month 12: number analyzed (Participants) | 36 | 26 | 13
  CD8-TNF-α [HPV-18], At Month 12 | 28.0 [7.0 to 101.0] | 18.0 [7.0 to 68.0] | 7.0 [7.0 to 7.0]

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms were assessed within 7 days post-vaccination. Unsolicited symptoms were assessed within 30 days post-vaccination. SAEs were assessed during the whole study period (from Day 0 up to Month 12).
Arm/Group | HIV+/Cervarix Group | HIV+/Aluminium Hydroxide Group | HIV-/Cervarix Group
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/59 | 0/30
Serious Adverse Events (participants affected / at risk) | 3/61 | 2/59 | 1/30
Other Adverse Events (participants affected / at risk) | 61/61 | 55/59 | 29/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV+/Cervarix Group (N=61) | HIV+/Aluminium Hydroxide Group (N=59) | HIV-/Cervarix Group (N=30)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — up to Month 12
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — up to Month 12
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — up to Month 12
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) — up to Month 12
Psychotic disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — up to Month 12
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) — up to Month 12
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) — up to Month 12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV+/Cervarix Group (N=61) | HIV+/Aluminium Hydroxide Group (N=59) | HIV-/Cervarix Group (N=30)
Pain (General disorders) | 52 (102) | 27 (36) | 28 (59)
Swelling (General disorders) | 19 (23) | 2 (2) | 12 (15)
Fatigue (General disorders) | 18 (20) | 16 (20) | 8 (15)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Acute stress disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5) | 2 (2)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 3 (3)
Bartholin's abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (3) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cd4 lymphocytes decreased (Investigations) | 2 (2) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 5 (5) | 4 (4)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 6 (7) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 4 (5) | 2 (3)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 2 (2) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 15 (18) | 11 (11) | 13 (19)
Headache (Nervous system disorders) | 31 (40) | 33 (48) | 18 (25)
Herpes simplex (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Herpes virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 7 (8) | 1 (1) | 4 (6)
Injection site induration (General disorders) | 4 (4) | 0 (0) | 4 (4)
Injection site mass (General disorders) | 3 (3) | 0 (0) | 0 (0)
Injection site pruritus (General disorders) | 3 (3) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Measles (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 2 (2) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4) | 7 (8)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 6 (6) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (2) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 3 (3) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 3 (3)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 1 (1) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 10 (11) | 10 (10) | 7 (7)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 2 (2)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 5 (5) | 4 (4) | 0 (0)
Vulvovaginal human papilloma virus infection (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 1 (1)
Vulvovaginitis trichomonal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.